Original Protocol and Amendments

March 8, 2018 - May 29, 2018

NCT04821245

ID: BRI IRB18-008

Defining Normal Postoperative Magnetic Resonance Imaging after Total Knee Arthroplasty

### Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: March 23, 2021

| Personnel Information | 1 |
|-----------------------------------------------------|----|
| Subject Checklist | 3 |
| Study Location | 4 |
| General Checklist | |
| Funding | 5 |
| Application Type Checklist | 6 |
| Expedited Paragraphs | 6 |
| Summary, Purpose, Procedures | 88 |
| Background and additional procedures | 9 |
| Subject Population | 10 |
| Recruitment Process, Subject Compensation and Costs | 11 |
| Risks | 13 |
| Benefits | 14 |
| Confidentiality | 14 |
| Consent Information | 16 |
| Assent Background | 17 |
| HIPAA | 18 |
| Drugs and Devices | 20 |
| Potential Conflict of Interest | 21 |
| Attachments | 21 |
| Obligations | 22 |

Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: March 23, 2021

| <b>Event Histor</b> | ry | .23 | 3 |
|---------------------|----|-----|---|
|---------------------|----|-----|---|

Protocol: IRB18-008 PI Name: Neal, Joseph Date Printed: March 23, 2021

Defining Normal Postoperative Magnetic Resonance Imaging after Total **Protocol Title:** 

Knee Arthroplasty

Draft

**Date Submitted:** 

**Approval Period:** 

This Print View may not reflect all comments and contingencies for approval. **Important Note:** 

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

## \* \* \* Personnel Information \* \* \*

Click "Help" (upper right corner of screen) for guidance regarding who to include below (Key Personnel) and what CITI Training is needed. See the Clinical Research Glossary for definitions. Questions: Contact the Research **Protections Department** 

### Principal Investigator

Client defines "Investigator" as an individual who conducts a research study. If the study is conducted by a team of individuals, the Investigator is the responsible leader of the team. Degree (MD/PhD/BSN/etc.) Name of Principal Investigator\* Title MD Neal, Joseph ANESTHESIOLOGIST **Phone** Email\* Fax 206-223-6980 Joseph.Neal@virginiamason.org **Investigator Affiliation Check ALL** VM/BRI Department Mailstop that apply\* Anesthesiology VM personnel B2-AN **BRI** personnel Zip code Other 98101 **Training Details** No training data is available.

### Sub-Investigator(s)

| Sub-Investigator | Degree<br>(MD/PhD/BSN/etc.) | Title | Research Department |
|---|---|---|---|
| Blackmore, Craig | MD | RADIOLOGIST | Radiology MD Admin |
| Verdin, Peter | | ORTHOPEDIC<br>SURGEON | Orthopedics - Outpatient |

### Sub-Investigator(s)

Name of Sub-Investigator(s) Degree (MD/PhD/BSN/etc.) Title

Blackmore, Craig RADIOLOGIST

Email\* **Phone** Fax

Craig.Blackmore@virginiamason.org 206-223-6851

**Investigator Affiliation Check ALL** VM/BRI Department Mailstop

that apply\*

Radiology MD Admin R3-324 VM personnel

> **BRI** personnel Zip code 98101 Other

Role in Study Radiologist \_\_\_\_\_\_

Training Details

No training data is available.

Sub-Investigator(s)

Name of Sub-Investigator(s) Degree (MD/PhD/BSN/etc.) Title

Verdin, Peter MD ORTHOPEDIC SURGEON

Email\*PhoneFaxPeter.Verdin@virginiamason.org206-223-7530X6-ORTVM/BRI DepartmentInvestigator Affiliation Check ALLMailstop

that apply\*

Orthopedics - Outpatient X VM personnel

BRI personnel Zip code Other 98101

Role in Study

| Training Details | | | |
|---|---|---|---|
| Course | UserID | CourseCompletionDate | CourseExpirationDate |
| CITI Good Clinical<br>Practice | peter.verdin | 11/14/2016 3:34:28 PM | 11/14/2019 3:34:28 PM |

## **Study Coordinator**

| Study Coordinator Degree (MD/PhD/BSN/etc.) | | Title | Research Department |
|---|---|---|---|
| Neal, Joseph | MD | ANESTHESIOLOGIST | Anesthesiology |

## **Study Coordinator**

Name of Study Coordinator Degree (MD/PhD/BSN/etc.) Title

Neal, Joseph MD ANESTHESIOLOGIST

Email\* Phone Fax

Joseph.Neal@virginiamason.org 206-223-8822

VM/BRI Department Investigator AffiliationCheck ALL Mailstop

that apply\*

Anesthesiology X VM personnel B2-AN

BRI personnel Zip code
Other 98101

Training Details

No training data is available.

### Regulatory Contact (Primary IRB contact if not PI or Study Coordinator)

| Name of Regulatory Contact | Degree (MD/PhD/BSN/etc.) | Title |
|----------------------------|--------------------------|-------|
| Email* | Phone | Fax |

\_\_\_\_\_

| VM/BRI Department | Investigator Affiliation Che that apply* | ck ALL Mailstop |
|---|---|---|
| | VM personnel | |
| | BRI personnel | Zip code |
| | Other | |
| Training Details | | |
| | No training data is ava | ailable. |

Additional Personnel Information: (Use the area below if necessary to provide additional information regarding the personnel on this protocol)

Dr. Lauren Steffel, Puget Sound VA Health Services, will participate in manuscript writing and data analysis. She will have no contact with Virginia Mason subjects. The data that she will have access to will be de-identified with regard to subject PHI.

\_\_\_\_\_

\* \* \* Subject Checklist \* \* \*

### **Subject Checklist**

Select all that apply:

Retrospective medical records (e.g. Chart Review)

Tissue, blood, other specimens (e.g. repository)

- X Individuals with underlying medical conditions
- X Healthy individuals

Select all vulnerable groups:

Check all targeted or possibly included subjects. This also applies to retrospective chart reviews. Some groups (e.g. prisoners, pregnant women, or children) may require additional IRB oversight per federal regulations.

#### **Prisoners**

45CFR46 Subpart C (Should be excluded unless you know subject(s) will be "in prison" at the time of enrollment. Notify IRB immediately if a subject becomes incarcerated after enrollment. This population can not be reviewed exempt.)

Pregnant women

45CFR46 Subpart B

Females of childbearing potential

Children (under 18)

45CFR46 Subpart D

Persons incompetent to give consent (e.g., dementia, comatose, have legally authorized representative)

Economically/educationally disadvantaged.

**Illiterate** 

Non-English speaking

See: VM Interpreter Services

Are any other subjects outside of the above targeted or possibly included in this study?

١

Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: March 23, 2021

| | * * * Study Lo | <br>cation * * * | |
|---|---|---|---|
| y Location | | | |
| Click "add" and create a s | separate row in the table I | below for each unique VM / BF | RI study location. |
| VM Location | Other VM Location: | VM location Study<br>Activities | Other Activities |
| Main Campus Seattle -<br>Clinic / Hospital | | Blood draw, Informed consent discussion, Ongoing study visits, Screening visits, Specific procedures associated with the study | |
| VM/BRI Table | | | |
| Location | Main Campus Seattle - Clinic | / Hospital | |
| Activity | Blood draw,Informed covisits,Specific procedure | onsent discussion,Ongoing stu<br>es associated with the study | dy visits,Screening |
| Are there any locations o below. If no, proceed to | utside of VM / BRI that are the next section. | e involved in any way with this | study? If yes, explain |
| i. Are any outside lo<br>more information r | cations "engaged"with this<br>egarding engagement) | s research study? If yes, expla | ain: (click on "Help" for |
| conducted at outsi | de locations? If yes, desc<br>Record for engaged activi | nt (IRB of Record) for any study<br>ribe in the table below (click "a<br>ties outside of VM in the space | idd"). If no, confirm |

Select All That Apply: At least 1 box must be checked to proceed. If none are applicable contact the IRB at IRB@benaroyaresearch.org Use the attachment section to add separate documents or forms.

Y Protected Health Information (PHI) will be viewed, created, accessed, used, or disclosed by VM/BRI personnel or others. (Checking this box activates the HIPAA section)

Protocol: IRB18-008 PI Name: Neal, Joseph Date Printed: March 23, 2021

-----

## Questionnaire/Survey

Tissues or data to be stored for future research projects (e.g. registry or repository)

Tissues or data to be sent out of VM / BRI as part of a research agreement - Material Transfer Agreement (MTA)- Data Use Agreement (DUA)

X FDA regulated device (Investigational or otherwise)- This includes Humanitarian Use Devices (HUD)

FDA regulated drugs, reagents, or chemicals (Investigational or otherwise)

This study is or will be posted on ClinicalTrials.gov If checked, specify number:

Radioisotopes/radiation-producing machines, even if standard of care (Radiation Safety)

VM/BRI Institutional Biosafety Committee (IBC) Review Required- Clinical research involving recombinant and/or synthetic nucleic acid

Request to Rely on Another IRB - Please upload completed Request to Rely and associated documents in attachment section (This applies for Cooperative Review studies.)

IRB Authorization Agreement (IAA), Memorandum Of Understanding (MOU), etc.(attach in the Attachments section (This only applies to studies where the Client IRB is the "Reviewing" IRB).

X A stand-alone protocol already exists.

Checking this box doesn't reduce the number of questions you need to answer. However, you can be brief with your answers and include references to the stand-alone protocol (e.g. section, page #) for more information. Use the attachment section to include the stand-alone protocol with your submission.

\_\_\_\_\_

\* \* \* Funding \* \* \*

### Funding / Resources

1) Is there funding or other resources required for this project?

No means absolutely no internal or external funds, services, skills, or products (e.g., statistical services, database warehousing, free test article) are provided. If no, proceed to the next section.

If yes, Click "add" and create a separate row in the table below for each unique funding source.

### Funding / Resources Table

| Funding<br>Name | BRI Funding<br># | | Unrestricted<br>BRI Funds | | | Industry<br>Funding |
|---|---|---|---|---|---|---|
| Washington<br>State<br>Society of<br>Anesthesiol<br>ogists<br>Seafair<br>Grant<br>Award | Through VM<br>Foundation | N | N | N | Y | N |

Funding / Resources Table

.....

Name of Funding Entity Washington State Society of Anesthesiologists Seafair Grant

BRI Funding Number Through VM Foundation

BRI restricted funds?

BRI unrestricted funds?

N
Federal Grant funds?

Non-Profit Foundation?

Y
Industry Funding

\_\_\_\_\_

## \* \* \* Application Type Checklist \* \* \*

Please check one of the boxes below to determine how to move forward with your project. The US Office of Human Research Protections (OHRP) has created graphic aids to help with deciding if your research requires IRB oversight. In addition, please contact the BRI Research Protections Department with questions.

### Application type checklist

Not Human Subjects Research (This form is not currently available through eProtocol. Please click "https://www.benaroyaresearch.org/sites/default/files/Human%20Subjects%20Determination%20Form.doc" target=\_blankhere if applicable.)

**Exempt** 

X Expedited/Full Board (This includes Cooperative and Chart Reviews.)

Indicate what level of review you anticipate for this protocol:

Full Board (greater than minimal risk)

X Expedited (minimal risk)

"https://www.benaroyaresearch.org/our-research/clinical-research/for-investigators/starting-study/cooperative-trials" target=\_blankCooperative (approval by another IRB of record, regardless of risk level)

### \* \* \* Expedited Paragraphs \* \* \*

EXPEDITED REVIEW CATEGORIES If this is a FULL BOARD study, or COOPERATIVE (IRB of Record is not BRI), then proceed to next section.

For expedited review all aspects of the research must be: (1) Minimal Risk (2) Involve one or more categories listed below. Select all that apply (Click Help for more information):

- Clinical studies of drugs and medical devices only when condition (a) and (b) are met.
  - Research on drugs for which an investigational new drug application (21 CFR Part 312) is not required. (Note: Research on marketed drugs that significantly increases the risks or decreases the acceptability of the risks associated with the use of the product is not eligible for expedited review.)
  - b) Research on medical devices for which
    - i) An investigational device exemption application (21 CFR Part 812) is not required; or
    - ii) The medical device is cleared/approved for marketing and the medical device is being used in accordance with its cleared/approved labeling.
- X 2. Collection of blood samples by finger stick, heel stick, ear stick, or venipuncture as follows:
  - a) From healthy, non-pregnant adults who weigh at least 110 pounds. For these subjects, the

\_\_\_\_\_

- amounts drawn may not exceed 550 ml in an 8 week period and collection may not occur more frequently than 2 times per week; or
- b) From other adults and children, considering the age, weight, and health of the subjects, the collection procedure, the amount of blood to be collected, and the frequency with which it will be collected. For these subjects, the amount drawn may not exceed the lesser of 50 ml or 3 ml per kg in an 8 week period and collection may not occur more frequently than 2 times per week.
- Prospective collection of biological specimens for research purposes by non-invasive means.

#### **Examples:**

- a) Hair and nail clippings in a non-disfiguring manner.
- b) Deciduous teeth at time of exfoliation or if routine patient care indicates a need for extraction.
- c) Permanent teeth if routine patient care indicates a need for extraction.
- d) Excreta and external secretions (including sweat).
- Uncannulated saliva collected either in an unstimulated fashion or stimulated by chewing gumbase or wax or by applying a dilute citric solution to the tongue.
- f) Placenta removed at delivery.
- g) Amniotic fluid obtained at the time of rupture of the membrane prior to or during labor.
- h) Supra- and subgingival dental plaque and calculus, provided the collection procedure is not more invasive than routine prophylactic scaling of the teeth and the process is accomplished in accordance with accepted prophylactic techniques.
- i) Mucosal and skin cells collected by buccal scraping or swab, skin swab, or mouth washings.
- j) Sputum collected after saline mist nebulization.
- X 4. Collection of data through non-invasive procedures (not involving general anesthesia or sedation) routinely employed in clinical practice, excluding procedures involving x-rays or microwaves. Where medical devices are employed, they must be cleared/approved for marketing. (Studies intended to evaluate the safety and effectiveness of the medical device are not generally eligible for expedited review, including studies of cleared medical devices for new indications.)

## **Examples:**

- a) Physical sensors that are applied either to the surface of the body or at a distance and do not involve input of significant amounts of energy into the subject or an invasion of the subject's privacy.
- b) Weighing or testing sensory acuity.
- c) Magnetic resonance imaging.
- Electrocardiography, electroencephalography, thermography, detection of naturally occurring radioactivity, electroretinography, ultrasound, diagnostic infrared imaging, doppler blood flow, and echocardiography.
- e) Moderate exercise, muscular strength testing, body composition assessment, and flexibility testing where appropriate given the age, weight, and health of the individual.
- X 5. Research involving materials (data, documents, records, or specimen) that have been collected, or will be collected solely for non-research purposes (such as medical treatment or diagnosis). (NOTE: Some research in this paragraph may be exempt from the HHS regulations for the protection of human subjects. 45 CFR 46.101(b)(4). This listing refers only to research that is not exempt.)
  - 6. Collection of data from voice, video, digital, or image recordings made for research purposes.
  - 7. Research on individual or group characteristics or behavior (including, but not limited to, research on

Protocol: IRB18-008 PI Name: Neal, Joseph Date Printed: March 23, 2021

\_\_\_\_\_

perception, cognition, motivation, identity, language, communication, cultural beliefs or practices, and social behavior) or research employing survey, interview, oral history, focus group, program evaluation, human factors evaluation, or quality assurance methodologies. (NOTE: Some research in this category may be exempt from the HHS regulations for the protection of human subjects - 45 CFR 46.101(b)(2) and (b)(3). This listing refers only to research that is not exempt.)

\_\_\_\_\_

\* \* \* Summary, Purpose, Procedures \* \* \*

BRI Study ID Number - From the Clinical Research Program (e.g. CRP170XX)

CRP18023

Unit / Department - Administrative Oversight of Research

Defining Normal Postoperative Magnetic Resonance Imaging after Total Knee Arthroplasty

### 1. Summary

Provide a summary of the scope of work of this protocol.

Recent reports(1) describe sentinel cases of presumed local anesthetic-induced myotoxicity occurring after continuous adductor canal blocks (CACB) that were placed to provide analgesia after total knee arthroplasty (TKA). Crucial to the diagnosis, management, and eventual understanding of this newly described anesthetic complication is elucidating what constitutes normal postoperative magnetic resonance imaging (MRI) after TKA. A recent retrospective review of MRIs obtained for various indications within a week of TKA failed to identify a consistent pattern of MR findings that might have defined "normal MRI imaging" after TKA (BRI 16092, Magnetic Resonance Imaging of the Quadriceps Muscle After Total Knee Arthroplasty). The logical next step in this investigation would be to obtain MRIs in TKR patients just prior to hospital discharge after an otherwise normal postoperative course.

2. Purpose

Describe the purpose for the proposed project as well as the hypotheses/research questions to be examined.

This knowledge is crucial for proper diagnosis and further understanding of this sentinel complication.

## 3. Procedures

 a) Describe the activities/procedures to be conducted in chronological order (e.g. pull charts/data from Cerner, screening, interventions/interactions with subjects, data collection, photographing, audio and video recording, follow-up.)

-Patients of various age and sex that are scheduled for unilateral TKR will be approached by VM orthopedic surgeons to ascertain their willingness to volunteer for this study

-Identified patients will be consented for study participation by the PI at least 24 hours prior to their entry into the study
-All patients will undergo the standard VMMC TKA clinical pathway, which includes a 2 day continuous adductor canal block
-If their postoperative course has been normal, 10 volunteers will undergo unilateral thigh MRI prior to discharge home on the
morning of postoperative day 2. These patients will have pre- and post-op CPK and aldolase levels analyzed.
-Leg MRIs will be graded using a standardized checklist by a supervised radiology resident who is unaware of the study's purpose.

b) Explain who will conduct the procedures. Include where and when they will take place.

-MRIs will be obtained as scheduled cases at VMMC

-CPK and aldolase will be obtained and analyzed by VMMC laboratory

by a radiologist who is unaware of the study's purpose

- c) Will you be conducting procedures directly with patients? If yes, answer the questions below. If no (e.g. Y chart review only), proceed to question 4.0 Study Duration.
  - i) Are there any procedures considered experimental and outside standard of care or established practices at Virginia Mason, including follow-up procedures?

Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: March 23, 2021

\_\_\_\_\_\_

#### If yes, explain.

Lower extremity MRIs are standard, but are not a routine part of postoperative TKA care. CPK and aldolase analyses before and after TKA is non-standard.

ii) Will blinding be involved with this study?

Υ

If yes, explain.

-The interpreting radiologist will be blinded as to the study's purpose

iii) Will deception be used?

V

If yes, provide a rationale and describe debriefing procedures. Submit a debriefing script in attachments section.

iv) Will audio, photographs, or video taping of individuals occur?

Ν

If yes, describe and clarify what will become of the tapes/photographs (e.g., shown at scientific meetings, erased, etc.).

4. Study Duration

What is the anticipated start date and duration of the proposed study?

We plan to start immediately after IRB approval. We anticipate all 20 volunteers should be recruited and studied within a 3 month period

\_\_\_\_\_

\* \* \* Background and additional procedures \* \* \*

- Background and additional procedures
- a. Relevant Background: Discuss the present knowledge, appropriate literature and rationale for conducting the research.

Local anesthetics consistently induce myotoxicity in animal models and in up to 0.5% of humans after ophthalmic blocks, yet clinically apparent myotoxicity in patients undergoing peripheral nerve blocks was heretofore believed to be nearly non-existent. (2) This changed after introduction of continuous adductor canal blocks (ACB) at Virginia Mason Medical Center when 4 patients developed symptoms, MRI findings, and neurophysiologic testing compatible with local anesthetic-induced myotoxicity. In short order, other cases were reported from the Swedish Orthopedic Institute, 3 from retrospective analysis of other post-TKA MRIs obtained at Virginia Mason, and anecdotally from practices throughout the United States. These sentinel complications have resulted in major morbidity for the affected patients. After a normal early postoperative course, the patients rapidly developed flaccid quadriceps muscles and the inability to lift the operative lower extremity against gravity, with consequent halting of their rehabilitative trajectory. While fortunate patients recovered fully or nearly so after weeks to a few months as the unaffected myoblasts regenerated, less fortunate patients have never recovered to baseline.

Because non-ophthalmic myotoxicity has never been described to this degree in humans, little is known about its etiology, diagnosis, and treatment. Definitive diagnosis of myositis requires muscle biopsy, but this invasive and expensive intervention is unlikely to occur. All patients in our series had MRI signals consistent with edema and inflammation, consistent with myositis. However, the radiologic literature is silent with regard to what constitutes normal MRI findings immediately after TKA. Therefore, the MRI pathology that we observed, while clearly demonstrating inflammatory changes in the anterior compartment of the leg, could conceivably represent normal postoperative findings. We have attempted to study this question by retrospectively reviewing MRIs of patients who underwent leg MRI within a week of TKA. While we could identify several patients with clinical presentations consistent with undiagnosed myotoxicity, we were unable to confidently discern pathological findings versus 'normal' postoperative changes on limaging

b. If applicable, please describe statistical methods of the research and plans for analysis of the data (i.e. planned statistics, justification of sample size, etc.).

Observational convenience sample, therefore N/A

c. Are there any alternative treatments to participating in this research (e.g., standard of care treatment, etc.)?

Ν

If yes, describe. Any standard treatment that is being withheld must be disclosed. This information must be included in the consent form. N/A d. Can subjects receive alternative treatment outside of enrolling in this study? Will subjects be followed after their participation is complete? N e. If yes, explain why and describe how: Is this a cooperative study (e.g. UW, FHCRC is IRB of record)? f. (If yes, answer the questions below. If no, proceed to the next section. Click here for more information.) Has this study been approved by the IRB of record? (NOTE: BRI IRB cannot review any COOP study not currently approved by the IRB of record) If yes, when did the initial approval for this study occur? ii. Has this study undergone Continuing Review (CR) at the IRB of record? If yes, what are the current approval dates? iii. Will there be any costs to VM for study procedures (e.g. lab costs, etc.)? If yes, how will these costs be paid to VM? (e.g., direct billing to your grant, etc.) Will potential subjects from VM be approached? iv. (Note: Refer to Non-VM Investigator Patient Approach Procedures for the correct procedures.) If yes, describe how subjects will be approached and by whom. \* \* \* Subject Population \* \* \* 6. **Subject Population** Complete the projected subject enrollment information below:List multiple subject groups/cohorts as a) appropriate.(e.g. retrospective, prospective, children, adult, controls, treatment, etc.)

## **Subject Enrollment**

| Subject Group<br>(DEFINE:<br>cases/controls/records/<br>specimens etc.) | Age Range | Expected Number at End of Study (locally) | Expected Enrollment next 12 months |
|---|---|---|---|
| 20 | 50-75 | 20 | 20 |

b) Complete the vulnerable subject table below:

## Potentially Vulnerable Subject Populations

| | Targeted | Possible Inclusion | Excluded | N/A |
|---|---|---|---|---|
| Prisoners: FAQ (Note: should be excluded unless you know subjects will be "in prison" at the time of enrollment. Notify IRB immediately if a subject becomes incarcerated after enrollment.) | | | X | |
| Pregnant Women: (45CFR Subpart B) | | | X | |
| Children (under 18): 45CFR46 Subpart D | | | X | |
| People not competent to provide informed consent | | | X | |
| If the above populations are targeted or possibly included, explain: (Give rationale and specific steps to protect those populations) | | | | |
| Female of childbearing potential: | | | X | |
| If excluded, explain: | | | | |
| Non-English Speaking: VM Interpreter Services | | | X | |
| If Non-English Speaking subjects are targeted or possibly included, give rationale and specific steps to protect those populations. If excluded, explain. | translator that | this study involv<br>hat are not part | derstanding thro<br>es the acquisition<br>of a standard kr | on of MRI and |
| New Description | New<br>Description | New<br>Description | New<br>Description | New<br>Description |
| New Description | New<br>Description | New<br>Description | New<br>Description | |

- Are any other potentially vulnerable subjects (sight impaired, illiterate, etc.) targeted or possibly included N c) in this study? If yes, explain and provide steps to protect this population:
- Inclusion and Exclusion Criteria (e.g., Participants must have 20/20 vision, Participants must be 30-45 d) years of age, etc.)
  - i. Identify inclusion criteria.

-Anticipated unilateral TKA performed under the standard VMMC joint pathway, with 2 night stay postop -Subjects will be operated by a single surgeon (Dr. Verdin) to eliminate possible confounders related to surgical technique -Subjects must be willing to volunteer for MRI study and CPK and aldolase blood draws

ii. Identify exclusion criteria.

-Any contraindication to use of spinal anesthesia or adductor canal-based analgesia

-History of muscle wasting or related disease

-History of auto-immune disorders that may affect the musculature

-History of pre-existing neurologic condition affecting the lower extremities

-Allergy to radiologic contrast -Contraindications to MRI exam

To provide support for your projected enrollment goals, how many patients at VMMC do you anticipate would have met your eligibility criteria over the last 1-5 years? If NA or no numbers available, explain why and provide rationale to support your projections:

1000 per year

| _ | | | | | | |
|---|---|---|---|---|---|---|
| f۱ | How long d | lo vou anticipate | it will take to | complete | accrual for this | etudy2 |
| 1 <i>1</i> | I IOW IOITU U | o vou anticipate | IL WIII LANG LU | COLLIDIE | acciual ioi iilio | Stuuv: |

3 months

\_\_\_\_\_

| | * * * Recruitment Process, Sub | oject Compensation and Costs * * * |
|---|---|---|
| 7. | Recruitment Process: | |
| a) | Describe the step-by-step procedures for identifying and recruiting potential research subjects and/or requesting their data or specimens. | |
| | willingness to volunteer for this study | r unilateral TKA will be approached by Dr. Verdin to ascertain their ation by the PI (Dr. Neal) at least 24 hours prior to their surgery |
| b) | Identify who will contact prospective subjects. ( | (complete request for waiver of consent if applicable) |
| , | Joseph M. Neal, MD | |
| c) | Planned Subject Identification Methods: | |
| , | VM Medical Records / Chart Review | Direct Advertising |
| | From PI's own practice / department | Referrals |
| | Records | |
| | Specific registries, specify IRB#: | |
| | Outside Institution, please specify: | |
| | X Other, explain below: | |
| | From VMMC orthopedic surgical patients scheduled Dr. Verdin or his physician assistant. | for TKA. Initial willingness to participate in the study will be ascertained by |
| d) | Planned Recruitment Materials / Methods: | |
| | X Face to face interactions | Flyers / posters |
| | Phone Scripts | Letters to providers / schools / organizations |
| | Television ads | Newspaper ads |
| | Letters to prospective subjects | Radio ads |
| | Oral Scripts | PowerPoint presentations |
| | Internet ads / postings | Email |
| | X Other, please specify: | Phone conversation with PI |
| | NA | |
| | Attach ALL recruitment information in its final form. | form using the Attachments section of this IRB eProtocol |
| | See BRI IRB Recruitment Material Guidance. | |
| 8. | Subject Compensation and Costs: | |
| a) | Will subjects or their health care providers be reproducts? | equired to pay for any study related procedures or N |
| | i. If "Yes," explain. Max out of pocket? Ar insurance will not cover study-related pro- | re any funds available from the study if the subjects ocedures or products? |

b) Will subjects receive compensation in any manner for participation? If "Yes," complete the questions N below. If "No", skip to the next section.

 Will subjects receive monetary payment? If yes, describe payment schedule including per visit and total. \_\_\_\_\_

| ii. | Will any one payment be more than 40% of total compensation? If "Yes," explain and provide |
|---|---|
| | rationale. |

iii. Will other forms of compensation be provided? If yes, describe below.

Parking Voucher Gifts
Transportation Lodging

Gift card/certificate Other (describe below)

\_\_\_\_\_

\* \* \* Risks \* \* \*

9. Risks / Data Safety Oversight / Monitoring

(Click "Help" above for more information)

- a) Pl's evaluation of the overall level of Risk. (Please check one: minimal, or greater than minimal.) Minimal risk: The probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life, or during the performance of routine physical or psychological examinations or tests.
  - Minimal riskGreater than minimal risk
- b) Check all potential risks/side effects to subjects. Check only added potential risks/side effects that may occur to subjects from the research and not those that would occur if subjects were to receive standard treatment/procedures only. [Note: Virtually all research studies involve "breach of confidentiality" and "invasion of privacy" as potential risks since several entities may have access to research records (e.g., FDA, NIH, IRB, etc.). Risks must be consistent with the consent form and protocol.]

#### Risk / Side Effects

| Physical Harms | | /chological | Social Economical | |
|---|---|---|---|---|
| Minor Pain Discomfort Serious Injury Death | | Depression | Х | Breach of Confidentiality, resulting in: |
| | | Confusion | | Invasion of privacy |
| | | | | Potential loss of employment or insurability |
| | | Stress | | Potential criminal prosecution |
| Injury from invasive medical procedure | al | Guilt | | |
| Harm from possible side e from drugs | ffects | Loss of self-esteem | | None (only applicable if all data is stripped of all identifiers and not coded) |
| X Rare allergic reaction to radiologic contrast dye | С | Embarrassment | | |
| None | Х | Possible anxiety or claustrophobia during MRI exam | | |
| | | None | | |

c) Describe the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological counseling resources).

-Standard assessment of allergy or MRI-associated risk prior to MRI study

| | -Standard care during phlebotomy -Referral to psychological counseling if indicated |
|---|---|
| | Who will be monitoring the risks noted above to ensure the safety of subjects? |
| | X The Principal Investigator Describe your monitoring plan for reviewing interim results and/or safety<br>concerns during the study: |
| | -Contact with the volunteer prior to obtaining the MRI -Post-procedural contact (after MRI and blood draw) to ascertain any concerns -Contact information of PI will be made available to the volunteers |
| | A group representing the study sponsor State name of group and describe monitoring plan for reviewing interim results and/or safety concerns during the study: |
| | A Data Safety Monitoring Board (DSMB) State name of DSMB and describe procedures for submitting summary reports from the DSMB to the IRB: |
| | Other: |
| | If multi-site trial, are DSMB report(s) available for research already conducted?If yes, attach DSMB reports. (see clinical research glossary for "DSMB" clarification. If you think your study warrants DSMB oversight and you do not know of one to utilize, please contact the IRB office.) |
| | Are there any stopping rules based on the risks noted above, or other study criteria? If yes, describe below and include study endpoints. (Click "Help" above for more information.)/ |
| - | * * * Benefits * * * |
| | Benefits(This section is not enabled for exempt or cooperative studies)/ |
| | Are there any direct benefits to the research participants? Note: Direct benefit is a valued or desired outcome; an advantage (please do not include monetary inducement or compensation). If yes, please describe. |
| | Are there any anticipated benefits of this study to society, academic knowledge or both? If yes, please describe. |
| | The results of this study should define the effectiveness of MRI and/or CPK / aldolase as diagnostic tools in future patients with suspected local anesthetic-induced myotoxicity |
| | Suspected total different induced myotoxions |
| | Explain how the potential benefits justify the potential risks involved in participation in this research. |
| _ | Explain how the potential benefits justify the potential risks involved in participation in this research. For this previously unknown complication, new knowledge is critical for both understanding the proper diagnosis and for complication management. We have tried other routes to understand the diagnostic paradigm, to no avail. The low risk and inconvenience of postoperative MRI and CPK / aldolase studies will facilitate further knowledge related to this previously unknown complication. |
| _ | Explain how the potential benefits justify the potential risks involved in participation in this research. For this previously unknown complication, new knowledge is critical for both understanding the proper diagnosis and for complication management. We have tried other routes to understand the diagnostic paradigm, to no avail. The low risk and inconvenience of |

| | | | | | | Date Printed: March |
|---|---|---|---|---|---|---|
| | | | - | | | |
| X | Identifiable | | | | | |
| | Anonymous | | | | | |
| Х | De-identified | | | | | |
| | Coded | | | | | |
| pass | word protected, cert | tificate of co | onfidentiality, etc.). In | rclude : | sa | i. coding system, limited access,<br>feguards to protect against direct or<br>its (e.g. publications): |
| -CPk<br>-A pa<br>gene | <ul> <li>reports contain patient range</li> <li>resword-protected spread</li> <li>rated MRI standard read</li> </ul> | names and med<br>Isheet housed<br>ing and CPK le | on a VMMC password-pro | will be s<br>otected o | eei | n only by Dr. Neal and the patient's orthopedic team<br>nputer will be used to link MRN to radiologist- |
| -Sub | ject number, age, results | of MRI and en | zyme analysis, sex. No ot | ther iden | tifia | able information |
| c) Othe | er than study staff an<br>or data that identify | d BRI Regu<br>subjects (inc | ulatory & Compliance cluding coded data)? | , what | er | ntities will have access to research record |
| NIH | | Stud | dy Sponsor | | | Contracted monitor |
| FDA | | Pers | sonal physician | | X | None |
| | Other: (explain below | v) | | | | |
| l) How | will research data b | e recorded | ? | | | |
| Case r | eport forms | Ren<br>cent | note data entry (e.g.<br>tral database off site) | ) | X | Local database (e.g. Excel spreadsheet) |
| REDC | ap database | Pati | ent medical records | | | N/A |
| | other: (explain below | <u>') </u> | | | | |
| e) How | will research record | s be stored | locally? | | | |
| VMMC | /BRI server | X Inve | estigator's computer | | | Locked file cabinet |
| Locked | | N/A | | | | Other: (explain below) |
| | | | | | | · |
| ) How | will specimens be s | tored? | | | | |
| | Limited access refri | gerator / fre | ezer | Lock | ed | cabinet / office |
| X | N/A | | | Othe | r: ( | (explain below) |
| g) After | completion of this s | tudy, will yo | ou keep any data and | l/or spe | eci | mens for future research purposes? N |
| if<br>re<br>b | yes then answer the<br>etained (i.e., possible<br>e submitted for addi | e following of<br>e use for an<br>tional use o | questions:Describe wother research projections fretained data and/c | hy the<br>ct[s], e<br>or speci | in<br>tc.<br>im | formation and/or specimens will be<br>). Note: Separate IRB applications must<br>ens outside the approved protocol: |
| | escribe in two or the | ree sentenc | es how the confident | iality of | f th | ne retained information and/or specimens |

Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: March 23, 2021

Indicate the length of time research records and/or specimens will be kept before EITHER all h) identifiers/codes are removed OR the records and/or specimens are destroyed. Describe the procedures you will use.

Research records will be kept 1 year after publication of our results. After that, the spreadsheet will be turned over to BRI for archiving.

\* \* \* Consent Information \* \* \*

#### Consent Information

**Consent Instructions and Checklist Template Consent Forms and Guidance** 

Click "Add" to enter information in the "Informed Consent" table below. This includes translated consents and waivers of consent. Exempt Studies: This table is disabled. If a consent is used then attach in the a) attachment section. Chart review: If accessing medical charts without consent, a waiver of consent is required. Oral Consent: A waiver of signed consent is required. Subjects under 18 yrs old: Go to the next section. complete and attach assent information. Enter information in the Informed Consent table separately for each consent and/or waiver of consent.

#### Informed Consent Table

| Title | Consent Type |
|-----------------------------------------------------------|--------------|
| Clean Consent - Vers. 04.09.18 - IRB18-008 | Consent |
| IRB Stamped Approved Consent - Vers. 04.09.18 - IRB18-008 | Consent |

## **Informed Consent Table**

Title (e.g. main, screening, translated, oral,

information sheet, waiver request) \*

Consent

Consent Information Type\*

Consent Document\*

X Attachment Clean Consent - Vers. 04.09.18 -IRB18-008

Clean Consent - Vers. 04.09.18 - IRB18-008

Who will obtain subjects consent? (Check all that apply)

Principal Investigator

Co-Investigator

**Study Coordinator** 

Research assistant(s)

Other research staff

**Contracted Data Collection Firm** 

Other (please specify)

### Informed Consent Table

Title (e.g. main, screening, translated, oral, information sheet, waiver request) \*

Consent Information Type\*

Consent Document\*

IRB Stamped Approved Consent - Vers. 04.09.18 - IRB18-008

Consent

Χ Attachment IRB Stamped Approved Consent -Vers. 04.09.18 - IRB18-008

Protocol: IRB18-008 PI Name: Neal, Joseph Date Printed: March 23, 2021

-----

| < | Principal Investigator |
|---|---------------------------------|
| X | Co-Investigator |
| | Study Coordinator |
| | Research assistant(s) |
| | Other research staff |
| | Contracted Data Collection Firm |
| | Other (please specify) |

If consenting human subjects answer the questions below. If NOT consenting human subjects, leave blank and skip to the next section.

b) Describe the process used to consent all subjects on the study.

-Volunteer subjects will be identified in orthopedic office by Dr. Verdin or his staff
-Those interested in participating will be consented by Joseph M. Neal, MD at least 24 hours prior to their surgery. If possible, consent will be obtained in person. If not possible, consent will be obtained via phone.

- c) Will subjects have as much time as they want between the explanation of the study and signing the consent form? If no, or N/A explain below.
- d) If consent is being obtained from non-English speaking subjects, explain the translation process for all documents seen by subjects, including consent documents. Describe the consent process in these circumstances.

N/A

- e) Do you plan on having a Legally Authorized Representative (LAR) involved in the consent process? If Nyes, explain below and ensure the appropriate section is included in the consent form.
- f) Will you require an impartial third party witness be included in the consenting process? If yes, explain below and ensure the appropriate section is included in the consent form.

-----

## \* \* \* Assent Background \* \* \*

- 13. Assent Background (Continue to the next section if no subjects under the age of 18 will be enrolled in this study)
- a) Complete the "Assent" table below. Attach assent documents and/or request assent waivers. Click "Help" above for more information regarding assent and assent waiver.

You must check children (under 18) on the Subject Checklist section to activate this table.

b) Complete the Regulatory Compliance worksheet below:

Regulatory Compliance - Subpart D - Children

Provide the specific age range for children (less than 18 years old) you wish to enroll in the study and what is

\_\_\_\_\_

| your accrual goal: | | | |
|---|---|---|---|
| Age Range: | | Total Accrual<br>Goal: | |
| Check the appropried CFR 46 subpart D | riate box below (only one) to indicate v<br>for research involving children. Chlic | vhich category your<br>k on the links below | study may be approved in light of 45 of for guidance. |
| | Research not involving greater than r | ninimal risk. 45 CF | R 46.404 |
| | Research involving greater than minimal risk, but presenting the prospect of direct benefit to the individual subjects. CFR 46.405 | | |
| | Research involving greater than minimal risk and no prospect of direct benefit to the individual child subjects involved in the research, but likely to yield generalizable knowledge about the subject's disorder or condition. 45 CFR 46.406 | | |
| | Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of children. 45 CFR 46.407 | | |
| | Will you be using an Assent Form? (-see 45 CFR 46.408 for reference) | Required for subjec | cts 7-11 years old per BRI IRB policies |
| approach(es) to su | Describe in the space below the details of your assent process for children in your study. (Include specific approach(es) to subjects in various age ranges, how assent will be documented, who will be able to give persimssion for each child (e.g. child's parent(s) or guardian), and how this permission will be recorded in the | | |
| | Does your study involve an FDA regulated drug, device, or biologic? If yes, check the appropriate box below (only one) to indicate which category your study may be approved in light of 21 CFR 50 Subpart D for research involving children. Click on the links below for guidance. | | |
| | Clinical investigations not involving g | reater than minimal | risk 21 CFR 50.51 |
| | Clinical investigations involving greater than minimal risk, but presenting the prospect of direct benefit to the individual subjects. 21 CFR 50.52 | | |
| | Clinical investigations involving greater than minimal risk and no prospect of direct benefit to individual subjects. | | |
| | Clinical investigations not otherwise a prevent, or alleviate a serious probler 50.53 | approvable that pres<br>maffecting the heal | sent an opportunity to understand,<br>th or welfare of children. 21 CFR |
| | Will you be using an Assent Form? ( - see 45 CFR 46.408 for reference) | Required for subject | cts 7-11 years old per BRI IRB policies |

\_\_\_\_\_\_

## \* \* \* HIPAA \* \* \*

14. Health Insurance Portability and Accountability Act (HIPAA)

If you are using PHI and this page is not active you must return to the General Checklist and check the box regarding the use of PHI in this research.

HIPAA Privacy Rule: Establishes the right of an individual to authorize a covered entity, such as health plan, health care clearinghouse or health care provider, to use and disclose his/her Protected Health Information (PHI) for research purposes. The Privacy Rule defines the elements of individual information that comprise PHI and establishes the conditions under which PHI may be used or disclosed by covered entities for research purposes. It also includes provisions to allow an individual's PHI to be disclosed or used in research without the person's authorization (i.e., IRB Waiver of HIPAA Requirement Authorization). For more information refer to the HIPAA Privacy Rule.

\_\_\_\_\_

Protected Health Information (PHI):Health information with one or more of the identifiers listed below. For more information see the NIH website. Research which involves the use of de-identified data is exempt from HIPAA requirements. In order to be de-identified data NONE of the subject identifiers listed below can be collected, used, reviewed, recoded, accessed or disclosed.

For more information see the following:VM/BRI Protected Health Information Guidance Document

- a) How will you obtain approval to access PHI for this research?
  - X HIPAA Authorization request from subject
    - X Incorporated into consent form

Stand alone document

Waiver of Subject HIPAA Authorization (partial or complete)(complete question e. below)

Limited Data Set and Data Use Agreement

Other: (explain below)

c) Will any non-VM/BRI personnel need access to PHI? If yes, how and where will they access subject PHI (e.g. on-site, remote via Cerner, etc.)?

d) Review the following list and indicate if any of the information will be collected from any medical records for the purpose of this research project.

**Names** 

**Social Security Numbers** 

**Telephone Numbers** 

All geographic subdivisions smaller than a state, including street address, city, county, precinct, zip code, and their equivalent geocodes, except for the initial three digits of a zip code, if according to the current publicly available data from the Bureau of the Census;

- The geographic unit formed by combining all zip codes with the same three initial digits contains more than 20,000 people; and
- ii. The initial three digits of a zip code for all such geographic units containing 20,000 or fewer people is changed to 000.

All elements of dates (except year) for dates directly related to an individual, including birth date, admission date, discharge date, date of death; and all ages over 89 and all elements of dates (including year) indicative of such age, except that such ages and elements may be aggregated into a single category of age 90 or older.

Fax Numbers

Electronic Mail Addresses (email)

- X Medical Record Numbers
  - i. You must identify the data points being collected from MRN by attaching a separate data collection sheet or listing them in the procedures section.

Health Plan Beneficiary Numbers

**Account Numbers** 

Certificate/License Numbers

Vehicle Identifiers and Serial Numbers, including License Plate Numbers

**Device Identifiers and Serial Numbers** 

Web Universal Resource Locations (URLs)

Internet Protocol (IP) Address Numbers

Biometric Identifiers, including Finger and Voice Prints

Full Face Photographic Images and any Comparable Images

Any other unique identifying number, character, or code (note this does not mean the unique code

assigned by the Investigator(s) to code the research data) Ν Are you requesting a HIPAA waiver? (Required for any type of waiver of consent) If yes, answer the e) following questions. If no, proceed to the next section. Explain why the research cannot reasonably be conducted without the waiver of authorization: ii. Explain why the research cannot reasonably be conducted without access to and use of identifiable health information: iii. Describe the reasonable safeguards to protect idenifiable information from unauthorized use or re-disclosure: iv. Describe the reasonable safeguards to protect against identification, directly or indirectly, any patient in any report of the research: Describe the plan to destroy the identifiers at the earliest opportunity consistent with the V. research. If there is a health or research justification for retaining identifiers, or if law requires you to keep such identifying information, please provide this information as well: vi. Provide written assurance that identifiable information will not be reused/disclosed to any other person or entity, unless such use is required by law, for oversight of the research study, or for other research permitted by law: Explain why the research is of sufficient importance to outweigh the privacy intrusion: vii. Explain who the subject should contact to enforce patient rights, or to obtain an accounting of viii. the research disclosures (e.g. Pl, sub-investigator, coordinator):

## \* \* \* Drugs and Devices \* \* \*

- **Drugs and Devices** 15.
- Does this study involve a drug or device? If YES, continue below.If NO, proceed to the next section. a)
  - Is the drug(s) or device(s) FDA approved? If YES, list drug / device name and explain in text

field below. (e.g. HDE, 510K, Compassionate Use, etc) If NO, click "add" and complete the table below for each investigational drug(s) or device(s).

MRI

(These tables are not activated unless a drug / device question is checked on the General Checklist section)

Briefly describe the drugs and devices listed above. Include any relevant information that has not been

\_\_\_\_\_\_

| described in the | he protocol | summary or | background | sections. |
|------------------|-------------|------------|------------|-----------|
|------------------|-------------|------------|------------|-----------|

MRI will be used to obtain thigh scans

\_\_\_\_\_

#### \* \* \* Potential Conflict of Interest \* \* \*

- Potential Conflict of Interest(This section is not enabled for exempt studies)/
- a) Y Is there funding for this study?
- b) N If yes, are there any positive financial disclosures related to this study for any key personnel?
- c) N Regardless of funding, are there any positive positional disclosures related to this study for any key personnel?
- d) Y I attest that I have read the 'https://brinet.benaroyaresearch.org/center/Documents/VM%20Research%20Conflicts%20of%20Interes t.pdf#search=research%20conflict'target='blank'VM Conflict of Interest Policy and agree to abide by its terms. I will update this protocol when new or changes in conflict of interest arise, and I will comply with any conflict management plan required by the Institutional Review Board (IRB) to manage, reduce, or eliminate any actual or potential conflict of interest for the duration of the research.

If Yes to b) or c) above, complete the table and answer the questions below concerning the potential conflict of interest. If No, then proceed to the next section.

Minimizing Risks and Disclosure to Subjects

- N Have you disclosed any actual, potential or perceived conflicts of interest in the consent form? Research
  Personnel are required to disclose all such conflicts to all research participants in the research consent
  form.
- f) What steps, if any, have you taken or will you take to manage the conflict of interest and minimize the risks associated with any actual, potential or perceived conflicts of interest arising out of this research?

\* \* \* Attachments \* \* \*

#### 16. Attachments

Attach relevant documents here. These could include:

- Collaborating Investigator's IRB approval and approved documents
- Conflict of Interest information
- Debriefing Script; Grant/Sub-contract
- HIPAA Authorization Form from HIPAA-covered entity
- Interview/Focus Group Questions
- Investigator's Brochure
- Letters of Agreement/Cooperation from organizations who will help with recruitment
- Questionnaires/Surveys
- Radiation Control Office approval material
- Recruitment Material (e.g., flyers, email text, verbal scripts)
- Protocol
- Patient Card
- Other files associated with the protocol (you can upload most standard file formats: xls, pdf, jpg, tif,

Protocol: IRB18-008 PI Name: Neal, Joseph Date Printed: March 23, 2021

\_\_\_\_\_

etc.)

Please be sure to attach all documents associated with your protocol. Failure to attach the necessary files may result in this protocol being returned prior to review.

To update or revise any attachments, please delete the existing attachment and upload the revised document to replace it.

| Select from list | Attachment Name | Attached Date | Submitted Date |
|---|---|---|---|
| Data Collection Sheet | IRB18-008 Copy of Study<br>Data Sheet | 03/08/2018 | |
| Other | IRB18-008 Neal Financial Disclosure | 03/08/2018 | |
| Data Collection Sheet | IRB18-008 Copy of MRI<br>Data Sheet | 03/08/2018 | |
| Protocol | Clean Protocol - Vers.<br>04.09.18 - IRB18-008 | 04/13/2018 | 04/13/2018 |

\_\_\_\_\_\_

## \* \* \* Obligations \* \* \*

Note: The use of "I" below refers to the Principal Investigator (PI). If someone other than the PI is completing and submitting this application, that person is responsible to make sure the PI is aware of their obligation and assurances cited below. The PI is ultimately responsible for all conduct under this study and answers provided in this IRB submission.

#### Research Obligations of the Principal Investigator Include the Following:

Training - ALL key personnel, including any newly added personnel, must meet all IRB required training requirements (e.g. CITI Ethics, GCP, Conflict of Interest). Training refreshers must be completed at the appropriate intervals (i.e. every three (3) or four (4) years).

Study Modifications - Changes to any aspect of the study (e.g. protocol, consent/assent forms, advertising materials, additional key personnel, subject population, etc.) will be submitted to the IRB for approval before instituting the changes.

Final Report - The IRB will be notified when the study is complete, and must be closed out in eProtocol prior to expiration of the approval.

#### Investigator's Statement and Assurance of Confidentiality:

I certify that I have reviewed this application, including attachments, and all information contained herein is accurate to the best of my knowledge.

I agree to not enroll any subject(s) or collect any data intended only for research use prior to issuance of an IRB approval.

I understand that I am fully responsible for the execution and management of this study, and I am responsible for the performance of any sub-investigators or key personnel, including their adherence to all of the applicable policies and regulations.

I agree to report any substantive changes to the information contained in this application, unanticipated problems, or adverse events encountered during the project immediately to the IRB.

I will ensure the names of any human subjects or any identifiable data from human subjects shall be treated as confidential information. This information will not be disclosed to anyone other than those directly connected with the research project unless the patient has given prior approval in writing.

If this is a funded project, I certify that the funding source document is entirely consistent with the corresponding study protocol.

I certify I have not been barred from doing research by any regulatory agency or entity. If I am a physician (or other licensed health care professional), I certify that my medical (or other) license is current.

I further agree any failure to perform the undertaking specified above shall be good cause for termination of the research project.

#### When Closing Your Protocol:

I understand when I close this protocol with the IRB NO further data collection, follow-up with subjects, coding of data, data analysis, and manuscript preparation that requires personal identifiable information (e.g. PHI) may be conducted.

I agree to retain all research materials for at least 10 years after closure of the research project and acknowledge these documents may be subject to review by the Clinical Research Program and IRB, if deemed necessary.

Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: March 23, 2021

I further certify I will not take any PHI and/or specimens generated from this research with me if I leave BRI/VM, unless having first established an agreement with VM legal in advance of my departure.

I confirm this study will not begin until the investigator receives written final approval or determination of exemption.

X The Principal Investigator has read and agrees to abide by the above obligations.

Continuing Review - You are responsible to complete and submit a Continuing Review form at least 30 days prior to the date of expiration. You will be asked to note accomplishments of your project at that time.

Protocol Deviations/Violations, Adverse Events (AEs) that occur in the course of the protocol will need to be submitted in a prompt manner from when they occurred.

X The Principal Investigator has read and agrees to abide by the above obligations.

Please click "next" to continue to protocol Check for Completeness. If the protocol is complete and ready for submission, please click "Submit Form" to your left to submit your protocol for IRB Review.

\_\_\_\_\_\_

## \* \* \* Event History \* \* \*

## **Event History**

| Date | Status | View Attachments | Letters |
|---|---|---|---|
| 05/07/2020 | CLOSED | | |
| 05/07/2020 | FINAL FORM<br>APPROVED | Υ | N |
| 04/27/2020 | PROTOCOL EXPIRED | | |
| 04/24/2020 | CONTINUING REVIEW 1<br>FORM Fox, Ellie added in<br>CONTINUING REVIEW | | |
| 04/23/2020 | FINAL FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 04/22/2020 | FINAL FORM<br>SUBMITTED | Υ | |
| 04/22/2020 | FINAL FORM CREATED | | |
| 05/30/2019 | CONTINUING REVIEW 1<br>FORM Stevens, Leslie<br>added in CONTINUING<br>REVIEW | | |
| 05/30/2019 | CONTINUING REVIEW 1<br>FORM Chan, Christine<br>added in CONTINUING<br>REVIEW | | |
| 04/25/2019 | CONTINUING REVIEW 1 FORM APPROVED | Υ | Υ |
| 04/22/2019 | CONTINUING REVIEW 1<br>FORM REVIEWER(S)<br>ASSIGNED | | |
| 04/19/2019 | CONTINUING REVIEW 1<br>FORM PANEL<br>MANAGER REVIEW | | |
| 04/19/2019 | CONTINUING REVIEW 1 FORM SUBMITTED | Υ | |

.....

| 04/19/2019 | CONTINUING REVIEW 1<br>FORM CREATED | | |
|------------|----------------------------------------------|---|---|
| 03/27/2019 | REPORT 1 FORM<br>WITHDRAWN | | |
| 03/27/2019 | REPORT 1 FORM<br>PANEL MANAGER<br>REVIEW | | |
| 03/22/2019 | REPORT 1 FORM<br>SUBMITTED | Y | |
| 03/13/2019 | AMENDMENT 3 FORM APPROVED | Y | Y |
| 03/01/2019 | SAE REPORT 1 FORM<br>APPROVED | Y | N |
| 03/01/2019 | AMENDMENT 3 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 03/01/2019 | SAE REPORT 1 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 03/01/2019 | AMENDMENT 3 FORM<br>PANEL MANAGER<br>REVIEW | | |
| 03/01/2019 | REPORT 1 FORM<br>CREATED | | |
| 03/01/2019 | SAE REPORT 1 FORM<br>SUBMITTED | Y | |
| 03/01/2019 | SAE REPORT 1 FORM<br>CREATED | | |
| 02/06/2019 | AMENDMENT 3 FORM SUBMITTED | Y | |
| 02/06/2019 | AMENDMENT 3 FORM CREATED | | |
| 05/31/2018 | AMENDMENT 2 FORM APPROVED | Υ | Y |
| 05/30/2018 | AMENDMENT 2 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 05/29/2018 | AMENDMENT 2 FORM SUBMITTED | Y | |
| 05/29/2018 | AMENDMENT 2 FORM CREATED | | |
| 05/24/2018 | AMENDMENT 1 FORM APPROVED | Y | Y |
| 05/23/2018 | AMENDMENT 1 FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 05/22/2018 | AMENDMENT 1 FORM SUBMITTED | Υ | |
| 05/17/2018 | AMENDMENT 1 FORM CREATED | | |
| 04/30/2018 | NEW FORM APPROVED | Υ | Y |

Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: March 23, 2021

| 04/30/2018 | NEW FORM UNDO<br>APPROVED | | |
|------------|-------------------------------------|---|---|
| 04/30/2018 | NEW FORM APPROVED | Υ | Υ |
| 04/17/2018 | NEW FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 04/13/2018 | NEW FORM<br>REVIEWER(S)<br>ASSIGNED | | |
| 04/12/2018 | NEW FORM PANEL<br>MANAGER REVIEW | | |
| 03/08/2018 | NEW FORM PANEL<br>ASSIGNED | | |
| 03/08/2018 | NEW FORM<br>SUBMITTED | Y | |



## NOTICE OF IRB EXEMPTION

Joseph Neal, MD Anesthesiology

RE: IRB# IRB18-008 (NEW)

Study Title: Defining Normal Postoperative Magnetic Resonance Imaging after Total Knee Arthroplasty

Dear Joseph Neal, MD,

Thank you for submitting the above referenced study for review by the Benaroya Research Institute at Virginia Mason Institutional Review Board (BRI IRB). Review was carried out in light of federal regulations on human subjects and BRI IRB policies.

During the course of the study, if there are changes in the protocol that would alter this determination (e.g. increased risk, additional non-exempt activity), including protocol termination, or if human subjects involved in the study are subjected to unanticipated problems, please report these immediately to BRI IRB. Please include the Protocol ID Number (IRB18-008) on all correspondence.

If your study received initial Feasibility Review, no study activity may occur until you receive a Clinical Research Program letter to commence from the BRI Administrative Director of Clinical Research, Cheryl Weaver. Her phone number is (206) 342-6911.

Please contact the Research Protections Department at irb@benaroyaresearch.org if you have any question regarding your approval or the eProtocol system. Thank you.

Sincerely,

Bredfeldt, James, MD

IRB Chair

Items included with this submission are listed below under attachments:

#### **Attachments**

Clean Protocol - Vers. 04.09.18 - IRB18-008

Notes:

Additional approved documents: IRB Stamped Approved Consent - Vers. 04.09.18 - IRB18-008



#### FINAL AUTHORIZATION TO COMMENCE CLINICAL RESEARCH

Days

33

125

158

Feasibility Submission to Approval

IRB Submission to Commencement

Notification

Total

DATE: August 16, 2018

TO: Joseph Neal MD, Principal Investigator

Leslie Stevens, Dept. Manager Maria Prado, Study Coordinator

| $ED \cap M_1$ | Chamil | Woose | Administrative | Director |
|---------------|--------|---------|----------------|----------|
| FRUM: | Chervi | weaver. | Administrative | Director |

Sylvia Cooper, CRP Specialist

RE: CRP18023 / IRB18-008

TITLE: Defining Normal Postoperative Magnetic Resonance Imaging after Total Knee Arthroplasty

This correspondence is to inform you that BRI's Clinical Research Program Administration has the following required documentation in our file for the above mentioned clinical research study:

- 1. BRI Feasibility email approving submission of your study to the IRB
- 2. IRB approval for the conduct of this study

Please remember, by proceeding with this project you are agreeing to comply with all regulations, (Institutional, State, Local and Federal) for Principal Investigators, as well as, those that guide the ethical conduct of clinical research. Any proposed changes or amendments to the project must be authorized by the Institutional Review Board, before they may be implemented.

We expect that your trial will accrue in a timely fashion and look forward to reviewing enrollment activity within 60 days of this authorization.

Sincerely,

Cheryl Waver, CCRC, CCRA Administrative Director, CRP cweaver@benaroyaresearch.org

CC: Research Protections Department

Tina Lencioni, Contract Administrator

Johnson Kukundakwe, Clinical Research Accountant

CRP Quality Assurance Department

Gail Chumbley, CRP Financial Manager

Erica Lacaden, Billing Specialist

David Caldwell, Communications Specialist



Protocol: IRB18-008 PI Name: Neal, Joseph Date Printed: March 01, 2019

Protocol Title: Defining Normal Postoperative Magnetic Resonance Imaging after Total

Knee Arthroplasty

Date Submitted: Draft Approval Period: Draft

Important Note: This Print View may not reflect all comments and contingencies for approval.

Please check the comments section of the online protocol.

Questions that appear to not have been answered may not have been required

for this submission. Please see the system application for more details.

-----

\*\*\*

#### ADVERSE EVENT REPORT FORM

- 1. Is this adverse event unexpected (in terms of nature, severity, or frequency) given (a) the research procedures described in the protocol-related documents, such as the IRB-approved research protocol and informed consent document, or the Investigator Brochure; and (b) the characteristics of the subject population being studied?
- 2. Is this adverse event related or possibly related to participation in the research (possibly related means there is a reasonable possibility the incident, experience, or outcome may have been caused by the drugs, devices or procedures involved in the research)?
- 3. Does this adverse event suggest the research places subjects or others at a greater risk of harm (including physical, psychological, economic, or social harm) than was previously known or recognized?

(Note: "off-site" reports will not be accepted unless; (a) the event described is both serious and unexpected,(b) the report identifies all previous safety reports concerning similar adverse experiences,(c) the report analyzes the significance of the current adverse experience in light of the previous reports, and (d) the report outlines a corrective action plan. 21 CFR 312.32)

If you answered "NO" to any of the above questions STOP. You do not need to submit this event/report to the IRB unless all three above criteria are met.

- 4. What type of report is this?
  - X Initial Report

| Date of Initial Report: | 03/01/2019 |
|--------------------------------|------------|
| Follow up # | |
| Follow up complete Drug | |
| Device | |
| N/A [Name of test article(s)]: | |

5. Describe in you are reporting (e.g. Confusion, Vomiting, Hyponatremia, etc.):

Catheters used for continuous adductor canal block contain wire. According to the manufacturer's published information, these catheters are deemed "MRI Conditional", with low to no risk from heating during an MRI scan.

Our first subject had their MRI on February 22, 2019 and reported a mild sensation of heating at the catheter site. The MRI was aborted. The patient reported no harm.

Dr. Neal became aware of this issue on February 25, 2019. After consultation with Drs. Blackmore, Strodtbeck, Warren, and Macdonald, it was agreed that the adductor canal catheter will be removed in subsequent patient volunteers that are recruited for this study.

- 6. **Event Start date:** 02/22/2019
- 7. Date of Death (if applicable):
- 8. Participant Study Identifier: Number 6
- 9. Why do you consider this event unexpected?

The manufacturer does not report significant heating to be an issue with these catheters. Furthermore, these catheters have indeed been in place in some patients who underwent uneventful MRI studies at Virginia Mason.

Protocol: IRB18-008 PI Name: Neal, Joseph

**IRB Protocol** BENAROYA RESEARCH INSTITUTE
Virginia Mason Date Printed: March 01, 2019 10. Relationship to research: **Definite Probable** Possible (possibly related means there is a reasonable probability that the incident, experience, or outcome may have been caused by the drugs, devices or procedures involved in the research.) Why do you consider this event related or possibly related to participation in the research? Warming at the catheter site is consistent with MRI effects on metallic objects What changes do you propose to the consent form and/or the protocol in order to protect the rights, welfare and safety of the research subjects? If none are proposed, provide the rationale for why changes are not needed? 13. Where did the unanticipated Adverse Event occur? (i.e. on site or off site) If "ON SITE" (e.g. occurred to VM/BRI subject) where did the AE occur? (e.g. VM, BRI, at home etc.): VMMC 5th floor MRI scanner 14) Choose an adverse event category: Death Life-Threatening Disability Hospitalization Congenital Required Medically Other: (explain below) Important Event Anomaly intervention to prevent damage / impairment Because the patient reported heating, the MRI was terminated. The heating immediately dissipated and the patient reported no further harm. 2/25/19 15) Date the PI/study staff became aware of this event: 16) Description of event: As noted above Has this event been reported to all appropriate agencies as defined in the protocol, grant, contract, or clinical trial agreement? Check all that apply and provide date reported: N/A Sponsor: **Date Notified:** N/A FDA (if BRI/VM PI holds the IND/IDE): **Date Notified:** N/A Coordinating Center: **Date Notified:** 

18) Has this type of event been reported previously to the BRI IRB? If yes, explain. I am unaware of any previous reports

Do you consider the frequency higher than expected? If yes, explain.

The event was unexpected based on previous experience and manufacturer report. What is unclear is the precise intensity of the heating reported by the patient. It is possible that other patients have experienced similar sensations, but have not reported them.

20) Is this study closed to new accrual at VM (and its affiliated sites)?

Ν

Ν





Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: March 01, 2019

| | i. | If yes, is at least one (1) participant at VM (and/or its affiliated sites) still receiving study treatment/intervention? |
|---|---|---|
| 21) | complet<br>underlin | if "yes" you will need to also<br>te an amendment form and attach the revised protocol and/or consent form with all changes<br>ned? |





Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: May 29, 2018

| Amendment | |
|-----------------------------------------------------|----|
| Personnel Information | 2 |
| Subject Checklist | 5 |
| Study Location | 5 |
| General Checklist | 6 |
| Funding | 7 |
| Application Type Checklist | 8 |
| Expedited Paragraphs | 8 |
| Summary, Purpose, Procedures | 10 |
| Background and additional procedures | 11 |
| Subject Population | 12 |
| Recruitment Process, Subject Compensation and Costs | 13 |
| Risks | 15 |
| Benefits | 16 |
| Confidentiality | 16 |
| Consent Information | 18 |
| Assent Background | 20 |
| HIPAA | 21 |
| Drugs and Devices | 23 |
| Potential Conflict of Interest | 23 |





Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: May 29, 2018

| Attachments | 24 |
|---------------|----|
| Obligations | 25 |
| Event History | 26 |



**Protocol Title:** 

**Date Submitted:** 

## IRB Protocol

05/29/2018

Defining Normal Postoperative Magnetic Resonance Imaging after Total Knee Arthroplasty

Protocol: IRB18-008 PI Name: Neal,Joseph Date Printed: May 29, 2018

| | Approval Period: | Draft | | | |
|---|---|---|---|---|---|
| | Important Note: This Print View may not reflect all comments and contingencies for approval. Please check the comments section of the online protocol. Questions that appear to not have been answered may not have been required for this submission. Please see the system application for more details. | | | | |
| | | *** | * * | | |
| | Protocol Amendment 1) C<br>attachments.3) Electronica<br>Remember to click "Subm<br>(see help above). Answer | ally "sign" your applicat<br>it Form" so the IRB sta | ion by clicking the chec<br>ff will receive your requ | approved protocol including a<br>k box in the Obligations sec<br>est.5) For Cooperative studi<br>spective. | any<br>tion.4)<br>ies |
| 1. | Does this amendment char complete the table. If no, c | nge the status of your sontinue to question 2. | tudy?If yes, check one | of the boxes below and | N |
| Stud | dy Status Change | | | 1 | |
| | Temporary Closure to | Accrual | Date Effective: | | |
| | Reason: | | | | |
| | Permanent Closure to<br>Particpation/Intervent | o Accrual, Study<br>ion Continues | Date Effective: | | |
| | How many subjects w this site? | vere ever enrolled at | | | |
| | How many subjects a this site? | re still on treatment at | | | |
| | How many subjects (tenrolled in this study know)? | total of all sites) were<br>(if applicable and | | | |
| | Permanent Closure to<br>Term Follow-Up and/o<br>Collection/Analysis Contraction/Intervention/Intervention/ | or Data<br>ontinues (no active | Date Effective: | | |
| | How many subjects w this site? | vere ever enrolled at | | | |
| | How many subjects (tenrolled in this study know)? | total of all sites) were<br>(if applicable and | | | |
| 2. | Describe all changes being referencing attachments cit | escribe all changes being proposed including any modifications to the attached documents. (If ferencing attachments cite page numbers) | | | |
| | Inclusion of stipend for particip 2. | ants | | | |
| 3. | Will the requested modifications change the scope or research objectives (e.g. change in specific aims, N change from previously approved use of human subjects, etc.)? If yes, describe below. | | | | ns, N |
| 4. | Are any NEW potentially vu (e.g. children, pregnant wor | | g added as targeted or | possibly included in this stud | dy N |

If yes, define your new study population and provide steps to protect the population. (Update the assent section if children are being added.)


| Were | | Consent Form? (If no consent, c | or no changes check "No" and proceed to Y |
|---|---|---|---|
| lf yes,<br>check | , describe changes be<br>the appropriate box(e | low and provide justification rega<br>es) below. Once this modification<br>all subjects as indicated. | arding your plan to re-consent subjects. Then, n is approved, the IRB will hold the researcher |
| | on of stipend and modificat | | |
| | Re-consent not requi | red | |
| X | • | ects with modified consent form( | (s) |
| | Re-consent active pa | articipants at next visit | • • |
| | Re-consent all subje | cts including those who have cor | npleted the study |
| | Other: (explain) | | |
| Indica | te level of risk involve | d with the changes proposed. | |
| (If | level of risk has chang | ged, update the "Risk" section in | the protocol.) |
| | Increase | X No Change | Decreased |
| If this<br>than r | study was originally reminimal risk of harm to | eviewed Expedited, do you attest<br>subjects? See the Help section | t this project continues to present no more Y for more information. |
| If no | , your study may be re | viewed by the Full Board IRB. | |
| pproval Ir | ncludes | | |
| st of secti | ons (and questions) th | at have been changed/modified | |
| | | * * * Personnel Informatio | n * * * |
| TI Trainin | ' (upper right corner of<br>ng is needed. See the<br>Department | screen) for guidance regarding<br>Clinical Research Glossary for c | who to include below (Key Personnel) and what<br>definitions. Questions: Contact the Research |
| incipal In | vestigator | | |
| ient defin | es "Investigator" as ar | n individual who conducts a resea<br>he responsible leader of the tear | arch study. If the study is conducted by a team |
| | incipal Investigator* | Degree (MD/PhD/BSN/etc.) | |
| _ | | MD | ANESTHESIOLOGIST |
| al, Joseph | | | |
| al, Joseph | | Phone | Fax |
| mail* | Qvirginiamason.org | Phone 206-223-6980 | Fax |

| Name of Principal Investigator* | De | Degree (MD/PhD/BSN/etc.) | | Title |
|---|---|---|---|---|
| Neal, Joseph | ME | D | | ANESTHESIOLOGIST |
| Email* | Pr | ione | | Fax |
| Joseph.Neal@virginiamason.org | | 206-223-6980 | | |
| VM/BRI Department | | vestigator Affiliation (<br>at apply* | Check ALL | Mailstop |
| Anesthesiology | Х | VM personnel | | B2-AN |
| | | BRI personnel | | Zip code |
| | | Other | | 98101 |



## No training data is available.

## Sub-Investigator(s)

| Sub-Investigator | Degree<br>(MD/PhD/BSN/etc.) | Title | Research Department |
|---|---|---|---|
| Blackmore, Craig | MD | RADIOLOGIST | Radiology MD Admin |
| Verdin, Peter | MD | ORTHOPEDIC<br>SURGEON | Orthopedics - Outpatient |
| Jackson, Dane | MD | RESIDENT -<br>RADIOLOGY | Graduate Medical<br>Education |

## Sub-Investigator(s)

Name of Sub-Investigator(s) Degree (MD/PhD/BSN/etc.) Title

Blackmore, Craig MD RADIOLOGIST

Email\* Phone Fax

Craig.Blackmore@virginiamason.org 206-223-6851

VM/BRI Department Investigator Affiliation Check ALL Mailstop

that apply\*

Radiology MD Admin X VM personnel R3-324

BRI personnel Zip code
Other 98101

Role in Study Radiologist

## **Training Details**

No training data is available.

## Sub-Investigator(s)

Name of Sub-Investigator(s) Degree (MD/PhD/BSN/etc.) Title

Verdin, Peter MD ORTHOPEDIC SURGEON

Email\*PhoneFaxPeter.Verdin@virginiamason.org206-223-7530X6-ORTVM/BRI DepartmentInvestigator Affiliation Check ALLMailstop

that apply\*

Orthopedics - Outpatient X VM personnel

BRI personnel Zip code Other 98101

## Role in Study

| Training Details | J Details | | |
|---|---|---|---|
| Course | UserID | CourseCompletionDate | CourseExpirationDate |
| CITI Good Clinical<br>Practice | peter.verdin | 11/14/2016 3:34:28 PM | 11/14/2019 3:34:28 PM |
| Human Research | peter.verdin | 11/8/2015 4:18:51 PM | 11/7/2018 9:00:00 PM |

## Sub-Investigator(s)

Name of Sub-Investigator(s) Degree (MD/PhD/BSN/etc.) Title

Jackson, Dane MD RESIDENT - RADIOLOGY





Email\* Phone Fax

Dane.Jackson@virginiamason.org 206-583-6079

VM/BRI Department Investigator Affiliation Check ALL Mailstop

that apply\*

Graduate Medical Education X VM personnel

BRI personnel Zip code

Other

Role in Study Masked assessment of MRI results

| Training Details | | | |
|---|---|---|---|
| Course | UserID | CourseCompletionDate | CourseExpirationDate |
| CITI Good Clinical<br>Practice | dane.jackson | 10/21/2017 3:19:35 PM | 10/20/2020 3:19:35 PM |
| Human Research | dane.jackson | 10/20/2017 2:09:36 PM | 10/19/2020 2:09:36 PM |

## **Study Coordinator**

| Study Coordinator | Degree<br>(MD/PhD/BSN/etc.) | Title | Research Department |
|---|---|---|---|
| Neal, Joseph | MD | ANESTHESIOLOGIST | Anesthesiology |

## **Study Coordinator**

Name of Study Coordinator Degree (MD/PhD/BSN/etc.) Title

Neal, Joseph MD ANESTHESIOLOGIST

Email\* Phone Fax

Joseph.Neal@virginiamason.org 206-223-8822

VM/BRI Department Investigator AffiliationCheck ALL Mailstop

that apply\*

Anesthesiology X VM personnel B2-AN

BRI personnel Zip code Other 98101

Training Details

No training data is available.

## Regulatory Contact (Primary IRB contact if not PI or Study Coordinator)

| Name of Regulatory Contact | Degree (MD/PhD/BSN/e | tc.) Title |
|---|---|---|
| Email* | Phone | Fax |
| VM/BRI Department | Investigator Affiliation C that apply* | neck ALL Mailstop |
| | VM personnel | |
| | BRI personnel | Zip code |



| | Other Dataile |
|---|---|
| 1 15 | raining Details No training data is available. |
| | Additional Personnel Information: (Use the area below if necessary to provide additional information regarding the personnel on this protocol) |
| | Dr. Lauren Steffel, Puget Sound VA Health Services, will participate in manuscript writing and data analysis. She will have no contact with Virginia Mason subjects. The data that she will have access to will be de-identified with regard to subject PHI. |
| | with Virginia Mason subjects. The data that she will have access to will be desidentified with regard to subject 1111. |
| • | * * * Subject Checklist * * * |
| Sı. | ubject Checklist |
| | Select all that apply: |
| | Retrospective medical records (e.g. Chart Review) |
| | Tissue, blood, other specimens (e.g. repository) |
| Х | Individuals with underlying medical conditions |
| Х | Healthy individuals |
| | Select all vulnerable groups: |
| | Check all targeted or possibly included subjects. This also applies to retrospective chart reviews. Some groups (e.g. prisoners, pregnant women, or children) may require additional IRB oversight per |
| | federal regulations. |
| | Prisoners |
| | 45CFR46 Subpart C (Should be excluded unless you know subject(s) will be "in prison" at the time of enrollment. Notify IRB immediately if a subject becomes incarcerated after enrollment. This population |
| | can not be reviewed exempt.) |
| | Pregnant women |
| | 45CFR46 Subpart B |
| | Females of childbearing potential |
| | Children (under 18) 45CFR46 Subpart D |
| | Persons incompetent to give consent (e.g., dementia, comatose, have legally authorized representative) |
| | Economically/educationally disadvantaged. |
| | Illiterate |
| | Non-English speaking |
| | See: VM Interpreter Services |
| Ar | re any other subjects outside of the above targeted or possibly included in this study? |
| | yes, describe below: |



# \* \* \* Study Location \* \* \*

## **Study Location**

Click "add" and create a separate row in the table below for each unique VM / BRI study location.

#### VM/BRI Table

| VM Location | Other VM Location: | VM location Study<br>Activities | Other Activities |
|---|---|---|---|
| Main Campus Seattle -<br>Clinic / Hospital | | Blood draw, Informed consent discussion, Ongoing study visits, Screening visits, Specific procedures associated with the study | |

### VM/BRI Table

**Location** Main Campus Seattle - Clinic / Hospital

Activity Blood draw, Informed consent discussion, Ongoing study visits, Screening

visits, Specific procedures associated with the study

| 2) | Are there any locations outside of VM / BRI that are involved in any way with this study? If yes, explain | Ν |
|---|---|---|
| • | below. If no, proceed to the next section. | |

- i. Are any outside locations "engaged" with this research study? If yes, explain: (click on "Help" for Note information regarding engagement)
- ii. Will the BRI IRB be responsible for oversight (IRB of Record) for any study procedures Normal conducted at outside locations? If yes, describe in the table below (click "add"). If no, confirm who is the IRB of Record for engaged activities outside of VM in the space below and then proceed to the next section.

-----

## \* \* \* General Checklist \* \* \*

### **General Checklist**

Select All That Apply: At least 1 box must be checked to proceed. If none are applicable contact the IRB at IRB@benaroyaresearch.org Use the attachment section to add separate documents or forms.

X Protected Health Information (PHI) will be viewed, created, accessed, used, or disclosed by VM/BRI personnel or others. (Checking this box activates the HIPAA section)

Questionnaire/Survey

Tissues or data to be stored for future research projects (e.g. registry or repository)

Tissues or data to be sent out of VM / BRI as part of a research agreement - Material Transfer Agreement



(MTA)- Data Use Agreement (DUA)

X FDA regulated device (Investigational or otherwise)- This includes Humanitarian Use Devices (HUD)

FDA regulated drugs, reagents, or chemicals (Investigational or otherwise)

This study is or will be posted on ClinicalTrials.gov If checked, specify number:

Radioisotopes/radiation-producing machines, even if standard of care (Radiation Safety)

VM/BRI Institutional Biosafety Committee (IBC) Review Required- Clinical research involving recombinant and/or synthetic nucleic acid

Request to Rely on Another IRB - Please upload completed Request to Rely and associated documents in attachment section (This applies for Cooperative Review studies.)

IRB Authorization Agreement (IAA), Memorandum Of Understanding (MOU), etc.(attach in the Attachments section (This only applies to studies where the Client IRB is the "Reviewing" IRB).

X A stand-alone protocol already exists.

Checking this box doesn't reduce the number of questions you need to answer. However, you can be brief with your answers and include references to the stand-alone protocol (e.g. section, page #) for more information. Use the attachment section to include the stand-alone protocol with your submission.

\_\_\_\_\_

\* \* \* Funding \* \* \*

#### Funding / Resources

1) Is there funding or other resources required for this project?

No means absolutely no internal or external funds, services, skills, or products (e.g., statistical services, database warehousing, free test article) are provided. If no, proceed to the next section.

If yes, Click "add" and create a separate row in the table below for each unique funding source.

### Funding / Resources Table

| Funding<br>Name | BRI Funding<br># | | Unrestricted<br>BRI Funds | | | Industry<br>Funding |
|---|---|---|---|---|---|---|
| Washington<br>State<br>Society of<br>Anesthesiol<br>ogists<br>Seafair<br>Grant<br>Award | Through VM<br>Foundation | N | N | N | Y | Z |

#### Funding / Resources Table

Name of Funding Entity

Washington State Society of Anesthesiologists Seafair Grant Award

**BRI Funding Number** 

Through VM Foundation

BRI restricted funds?

N



BRI unrestricted funds?

Federal Grant funds?

Non-Profit Foundation?

Industry Funding

N

\_\_\_\_\_

# \* \* \* Application Type Checklist \* \* \*

Please check one of the boxes below to determine how to move forward with your project. The US Office of Human Research Protections (OHRP) has created graphic aids to help with deciding if your research requires IRB oversight. In addition, please contact the BRI Research Protections Department with questions.

## Application type checklist

Not Human Subjects Research (This form is not currently available through eProtocol. Please click "https://www.benaroyaresearch.org/sites/default/files/Human%20Subjects%20Determination%20Form.doc" target= blankhere if applicable.)

**Exempt** 

X Expedited/Full Board (This includes Cooperative and Chart Reviews.)

Indicate what level of review you anticipate for this protocol:

Full Board (greater than minimal risk)

X Expedited (minimal risk)

"https://www.benaroyaresearch.org/our-research/clinical-research/for-investigators/starting-study/cooperative-trials" target=\_blankCooperative (approval by another IRB of record, regardless of risk level)

-----

## \* \* \* Expedited Paragraphs \* \* \*

EXPEDITED REVIEW CATEGORIES If this is a FULL BOARD study, or COOPERATIVE (IRB of Record is not BRI), then proceed to next section.

For expedited review all aspects of the research must be: (1) Minimal Risk (2) Involve one or more categories listed below. Select all that apply (Click Help for more information):

- 1 Clinical studies of drugs and medical devices only when condition (a) and (b) are met.
  - a) Research on drugs for which an investigational new drug application (21 CFR Part 312) is not required. (Note: Research on marketed drugs that significantly increases the risks or decreases the acceptability of the risks associated with the use of the product is not eligible for expedited review.)
  - b) Research on medical devices for which
    - i) An investigational device exemption application (21 CFR Part 812) is not required; or
    - ii) The medical device is cleared/approved for marketing and the medical device is being used in accordance with its cleared/approved labeling.
- X 2. Collection of blood samples by finger stick, heel stick, ear stick, or venipuncture as follows:
  - a) From healthy, non-pregnant adults who weigh at least 110 pounds. For these subjects, the amounts drawn may not exceed 550 ml in an 8 week period and collection may not occur more frequently than 2 times per week; or
  - b) From other adults and children, considering the age, weight, and health of the subjects, the



collection procedure, the amount of blood to be collected, and the frequency with which it will be collected. For these subjects, the amount drawn may not exceed the lesser of 50 ml or 3 ml per kg in an 8 week period and collection may not occur more frequently than 2 times per week.

3. Prospective collection of biological specimens for research purposes by non-invasive means.

## **Examples:**

- a) Hair and nail clippings in a non-disfiguring manner.
- b) Deciduous teeth at time of exfoliation or if routine patient care indicates a need for extraction.
- c) Permanent teeth if routine patient care indicates a need for extraction.
- d) Excreta and external secretions (including sweat).
- e) Uncannulated saliva collected either in an unstimulated fashion or stimulated by chewing gumbase or wax or by applying a dilute citric solution to the tongue.
- f) Placenta removed at delivery.
- g) Amniotic fluid obtained at the time of rupture of the membrane prior to or during labor.
- h) Supra- and subgingival dental plaque and calculus, provided the collection procedure is not more invasive than routine prophylactic scaling of the teeth and the process is accomplished in accordance with accepted prophylactic techniques.
- i) Mucosal and skin cells collected by buccal scraping or swab, skin swab, or mouth washings.
- j) Sputum collected after saline mist nebulization.
- X 4. Collection of data through non-invasive procedures (not involving general anesthesia or sedation) routinely employed in clinical practice, excluding procedures involving x-rays or microwaves. Where medical devices are employed, they must be cleared/approved for marketing. (Studies intended to evaluate the safety and effectiveness of the medical device are not generally eligible for expedited review, including studies of cleared medical devices for new indications.)

## **Examples:**

- a) Physical sensors that are applied either to the surface of the body or at a distance and do not involve input of significant amounts of energy into the subject or an invasion of the subject's privacy.
- b) Weighing or testing sensory acuity.
- c) Magnetic resonance imaging.
- Electrocardiography, electroencephalography, thermography, detection of naturally occurring radioactivity, electroretinography, ultrasound, diagnostic infrared imaging, doppler blood flow, and echocardiography.
- e) Moderate exercise, muscular strength testing, body composition assessment, and flexibility testing where appropriate given the age, weight, and health of the individual.
- X 5. Research involving materials (data, documents, records, or specimen) that have been collected, or will be collected solely for non-research purposes (such as medical treatment or diagnosis). (NOTE: Some research in this paragraph may be exempt from the HHS regulations for the protection of human subjects. 45 CFR 46.101(b)(4). This listing refers only to research that is not exempt.)
  - 6. Collection of data from voice, video, digital, or image recordings made for research purposes.
  - 7. Research on individual or group characteristics or behavior (including, but not limited to, research on perception, cognition, motivation, identity, language, communication, cultural beliefs or practices, and social behavior) or research employing survey, interview, oral history, focus group, program evaluation, human factors evaluation, or quality assurance methodologies. (NOTE: Some research in this category



| may be exempt from the HHS regulations for the protection of humand (b)(3). This listing refers only to research that is not exempt.) | an subjects - 45 CFR 46.101(b)(2 |
|---|---|
| * * * Summary, Purpose, Procedures * * | * |
| BRI Study ID Number - From the Clinical Research Program (e.g. RP170XX) | CRP18023 |

## 1. Summary

Provide a summary of the scope of work of this protocol.

Recent reports(1) describe sentinel cases of presumed local anesthetic-induced myotoxicity occurring after continuous adductor canal blocks (CACB) that were placed to provide analgesia after total knee arthroplasty (TKA). Crucial to the diagnosis, management, and eventual understanding of this newly described anesthetic complication is elucidating what constitutes normal postoperative magnetic resonance imaging (MRI) after TKA. A recent retrospective review of MRIs obtained for various indications within a week of TKA failed to identify a consistent pattern of MR findings that might have defined "normal MRI imaging" after TKA (BRI 16092, Magnetic Resonance Imaging of the Quadriceps Muscle After Total Knee Arthroplasty). The logical next step in this investigation would be to obtain MRIs in TKR patients just prior to hospital discharge after an otherwise normal postoperative course.

### 2. Purpose

Describe the purpose for the proposed project as well as the hypotheses/research questions to be examined.

This study aims to define normal quadriceps imaging in 20 asymptomatic volunteers one to two days after undergoing TKA. A secondary aim is to investigate alterations in creatine phosphokinase (CPK) and aldolase levels coincident with TKA. The aim of this observational study is to define what constitutes a normal MRI appearance and normal CPK / aldolase alterations in postoperative TKA patients. This knowledge is crucial for proper diagnosis and further understanding of this sentinel complication.

### 3. Procedures

 a) Describe the activities/procedures to be conducted in chronological order (e.g. pull charts/data from Cerner, screening, interventions/interactions with subjects, data collection, photographing, audio and video recording, follow-up.)

-Patients of various age and sex that are scheduled for unilateral TKR will be approached by VM orthopedic surgeons to ascertain their willingness to volunteer for this study

-identified patients will be consented for study participation by the PI at least 24 hours prior to their entry into the study -All patients will undergo the standard VMMC TKA clinical pathway, which includes a 1 to 2 day continuous adductor canal block

-If their postoperative course has been normal,

These patients will have pre- and post-op CPK and aldolase

levels analyzed.

-Leg MRIs will be graded using a standardized checklist by a supervised radiology resident who is unaware of the study's purpose.

b) Explain who will conduct the procedures. Include where and when they will take place.

-MRIs will be obtained as scheduled cases at VMMC

-CPK and aldolase will be obtained and analyzed by VMMC laboratory

-MRIs will be assessed using a standardize template by a radiologist who is unaware of the study's purpose

- c) Will you be conducting procedures directly with patients? If yes, answer the questions below. If no (e.g. Y chart review only), proceed to question 4.0 Study Duration.
  - i) Are there any procedures considered experimental and outside standard of care or established practices at Virginia Mason, including follow-up procedures?

If yes, explain.

Lower extremity MRIs are standard, but are not a routine part of postoperative TKA care. CPK and aldolase analyses before

N



ii)

-----

| and after TKA is non-standard. | |
|-------------------------------------------------------------------------|---|
| Will blinding be involved with this study? If yes, explain. | Υ |
| -The interpreting radiologist will be blinded as to the study's purpose | - |

iii) Will deception be used?

If yes, provide a rationale and describe debriefing procedures. Submit a debriefing script in attachments section.

iv) Will audio, photographs, or video taping of individuals occur?

If yes, describe and clarify what will become of the tapes/photographs (e.g., shown at scientific meetings, erased, etc.).

4. Study Duration

What is the anticipated start date and duration of the proposed study?

We plan to start immediately after IRB approval. We anticipate all 20 volunteers should be recruited and studied within a 3 month period

-----

\* \* \* Background and additional procedures \* \* \*

- Background and additional procedures
- a. Relevant Background: Discuss the present knowledge, appropriate literature and rationale for conducting the research.

Local anesthetics consistently induce myotoxicity in animal models and in up to 0.5% of humans after ophthalmic blocks, yet clinically apparent myotoxicity in patients undergoing peripheral nerve blocks was heretofore believed to be nearly non-existent. (2) This changed after introduction of continuous adductor canal blocks (ACB) at Virginia Mason Medical Center when 4 patients developed symptoms, MRI findings, and neurophysiologic testing compatible with local anesthetic-induced myotoxicity. In short order, other cases were reported from the Swedish Orthopedic Institute, 3 from retrospective analysis of other post-TKA MRIs obtained at Virginia Mason, and anecdotally from practices throughout the United States. These sentinel complications have resulted in major morbidity for the affected patients. After a normal early postoperative course, the patients rapidly developed flaccid quadriceps muscles and the inability to lift the operative lower extremity against gravity, with consequent halting of their rehabilitative trajectory. While fortunate patients recovered fully or nearly so after weeks to a few months as the unaffected myoblasts regenerated, less fortunate patients have never recovered to baseline.

Because non-ophthalmic myotoxicity has never been described to this degree in humans, little is known about its etiology, diagnosis, and treatment. Definitive diagnosis of myositis requires muscle biopsy, but this invasive and expensive intervention is unlikely to occur. All patients in our series had MRI signals consistent with edema and inflammation, consistent with myositis. However, the radiologic literature is silent with regard to what constitutes normal MRI findings immediately after TKA. Therefore, the MRI pathology that we observed, while clearly demonstrating inflammatory changes in the anterior compartment of the leg, could conceivably represent normal postoperative findings. We have attempted to study this question by retrospectively reviewing MRIs of patients who underwent leg MRI within a week of TKA. While we could identify several patients with clinical presentations consistent with undiagnosed myotoxicity, we were unable to confidently discern pathological findings versus 'normal' postoperative changes on imaging.

b. If applicable, please describe statistical methods of the research and plans for analysis of the data (i.e. planned statistics, justification of sample size, etc.).

Observational convenience sample, therefore N/A

c. Are there any alternative treatments to participating in this research (e.g., standard of care treatment, etc.)?

If yes, describe. Any standard treatment that is being withheld must be disclosed. This information must be included in the consent form.



| Can su | ubiects recei | ive alternative t | treatment outside of enro | olling in this study? | N/A |
|---|---|---|---|---|---|
| | Will subjects be followed after their participation is complete? | | | | |
| If yes, explain why and describe how: | | | | | |
| Is this | a cooperativ | ve study (e.g. U | JW, FHCRC is IRB of red | cord)? | N |
| (If yes, answer the questions below. If no, proceed to the next section. Click here for more information.) | | | | | |
| <ul> <li>Has this study been approved by the IRB of record? (NOTE: BRI IRB cannot review an<br/>COOP study not currently approved by the IRB of record)</li> </ul> | | | | | |
| | If yes, wh | en did the initia | al approval for this study | occur? | |
| ii. Has this study undergone Continuing Review (CR) at the IRB of record? | | | | | |
| If yes, what are the current approval dates? | | | | | |
| iii. Will there be any costs to VM for study procedures (e.g. lab costs, etc.)? | | | | | |
| | If yes, how will these costs be paid to VM? (e.g., direct billing to your grant, etc.) | | | | |
| iv. | ···· postantial conference of production | | | | |
| (Note: Refer to Non-VM Investigator Patient Approach Procedures for the correct procedures.) If yes, describe how subjects will be approached and by whom. | | | | | |
| | | | * * * Subject Population | n * * * | |
| Subjec | Subject Population | | | | |
| Comple | ete the proje<br>priate.(e.g. r | ected subject e<br>retrospective, p | nrollment information be<br>prospective, children, adu | low:List multiple subject g | groups/cohorts as<br>c.) |
| ject Enro | ollment | | | | |
| ject Grou<br>FINE:<br>es/contro | up<br>ols/records/ | Age Range | Expected Number at End of Study (locally) | Expected Number at End of Study (Total if multi-site) | Expected Enrollment next 12 months |

| (DEFINE: cases/controls/records/specimens etc.) | Age Range | End of Study (locally) | End of Study (Total if multi-site) | next 12 months |
|---|---|---|---|---|
| 20 | 50-75 | 20 | | 20 |

b) Complete the vulnerable subject table below:

Potentially Vulnerable Subject Populations



| | Targeted | Possible Inclusion | Excluded | N/A |
|---|---|---|---|---|
| Prisoners: FAQ (Note: should be excluded unless you know subjects will be "in prison" at the time of enrollment. Notify IRB immediately if a subject becomes incarcerated after enrollment.) | | | X | |
| Pregnant Women: (45CFR Subpart B) | | | X | |
| Children (under 18): 45CFR46 Subpart D | | | Χ | |
| People not competent to provide informed consent | | | Χ | |
| If the above populations are targeted or possibly included, explain: (Give rationale and specific steps to protect those populations) | | | | |
| Female of childbearing potential: | | | X | |
| If excluded, explain: | | | | |
| Non-English Speaking: VM Interpreter Services | | | Х | |
| If Non-English Speaking subjects are targeted or possibly included, give rationale and specific steps to protect those populations. If excluded, explain. | translator that | ding not fully un<br>this study involv<br>hat are not part<br>ospitalization | es the acquisition | on of MRI and |
| New Description | New<br>Description | New<br>Description | New<br>Description | New<br>Description |
| New Description | New<br>Description | New<br>Description | New<br>Description | |

- c) Are any other potentially vulnerable subjects (sight impaired, illiterate, etc.) targeted or possibly included N in this study? If yes, explain and provide steps to protect this population:
- d) Inclusion and Exclusion Criteria (e.g., Participants must have 20/20 vision, Participants must be 30-45 years of age, etc.)
  - i. Identify inclusion criteria.

-Anticipated unilateral TKA performed under the standard VMMC joint pathway, with 1 to 2 night stay postop -Subjects will be operated by a single surgeon (Dr. Verdin) to eliminate possible confounders related to surgical technique -Subjects must be willing to volunteer for MRI study and CPK and aldolase blood draws

ii. Identify exclusion criteria.

-Any contraindication to use of spinal anesthesia or adductor canal-based analgesia

-History of muscle wasting or related disease

-History of auto-immune disorders that may affect the musculature

-History of pre-existing neurologic condition affecting the lower extremities

-Allergy to radiologic contrast

-Contraindications to MRI exam

e) To provide support for your projected enrollment goals, how many patients at VMMC do you anticipate would have met your eligibility criteria over the last 1-5 years? If NA or no numbers available, explain why and provide rationale to support your projections:

1000 per year

| f) | How long do y | vou anticipate | it will take to | complete | accrual for | this study? |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

3 months

\_\_\_\_\_

<sup>\* \* \*</sup> Recruitment Process, Subject Compensation and Costs \* \* \*



| | Recrui | tment Process: | | |
|---|---|---|---|---|
| | Describe the step-by-step procedures for identifying and recruiting potential research subjects and/or requesting their data or specimens. | | | |
| | willi | tients of various age and sex that are scheduled for unila<br>ngness to volunteer for this study<br>ntified patients will be consented for study participation b | eral TKA will be approached by Dr. Verdin to ascertain their ythe PI (Dr. Neal) at least 24 hours prior to their surgery | |
| | | | elete request for waiver of consent if applicable) | |
| | Jose | eph M. Neal, MD | | |
| | Planne | ed Subject Identification Methods: | | |
| | VI | M Medical Records / Chart Review | Direct Advertising | |
| | Fr | rom PI's own practice / department | Referrals | |
| | Re | ecords | | |
| | S | pecific registries, specify IRB#: | | |
| | O | utside Institution, please specify: | | |
| | X O | ther, explain below: | | |
| | | rom VMMC orthopedic surgical patients scheduled for TK r. Verdin or his physician assistant. | A. Initial willingness to participate in the study will be ascertained | by |
| | Planne | ed Recruitment Materials / Methods: | | |
| | X Fa | ace to face interactions | Flyers / posters | |
| | Pl | none Scripts | Letters to providers / schools / organizations | |
| | Te | elevision ads | Newspaper ads | |
| | Le | etters to prospective subjects | Radio ads | |
| | O | ral Scripts | PowerPoint presentations | |
| | | ternet ads / postings | Email | |
| | X O | ther, please specify: | Phone conversation with PI | |
| | N | A | | |
| | Attacl form. | h ALL recruitment information in its final form | using the Attachments section of this IRB eProtocol | |
| | See E | BRI IRB Recruitment Material Guidance. | | |
| | Subjec | ct Compensation and Costs: | | |
| | Will su<br>produc | bjects or their health care providers be requirents? | ed to pay for any study related procedures or | N |
| | i. | If "Yes," explain. Max out of pocket? Are an insurance will not cover study-related proced | / funds available from the study if the subjects ures or products? | |
| , | Will su<br>below. | bjects receive compensation in any manner for If "No", skip to the next section. | or participation? If "Yes," complete the questions | Υ |
| | i. | Will subjects receive monetary payment? and total. | f yes, describe payment schedule including per visit | Υ |
| | \$50 | stipend will be paid after the participant has completed the | ne study (naid as gift card) | |



| <br> | <br> |
|------|------|

- ii. Will any one payment be more than 40% of total compensation? If "Yes," explain and provide rationale.
- ii. Will other forms of compensation be provided? If yes, describe below.

Υ

Parking Voucher

Gifts Lodging

Transportation

Lodging

X Gift card/certificate

Other (describe below)

As noted above

\* \* \* Risks \* \* \*

9. Risks / Data Safety Oversight / Monitoring

(Click "Help" above for more information)

- a) Pl's evaluation of the overall level of Risk. (Please check one: minimal, or greater than minimal.) Minimal risk: The probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life, or during the performance of routine physical or psychological examinations or tests.
  - X Minimal riskGreater than minimal risk
- b) Check all potential risks/side effects to subjects. Check only added potential risks/side effects that may occur to subjects from the research and not those that would occur if subjects were to receive standard treatment/procedures only. [Note: Virtually all research studies involve "breach of confidentiality" and "invasion of privacy" as potential risks since several entities may have access to research records (e.g., FDA, NIH, IRB, etc.). Risks must be consistent with the consent form and protocol.]

#### Risk / Side Effects

| Ph | Physical Harms | | ychological | So | cial Economical |
|---|---|---|---|---|---|
| | Minor Pain | | Depression | Х | Breach of Confidentiality, resulting in: |
| | Discomfort | | Confusion | Х | Invasion of privacy |
| | Serious Injury | | Hallucination | | Potential loss of employment or insurability |
| | Death | | Stress | | Potential criminal prosecution |
| | Injury from invasive medical procedure | | Guilt | | |
| | Harm from possible side effects from drugs | | Loss of self-esteem | | None (only applicable if all data is stripped of all identifiers and not coded) |
| Х | Rare allergic reaction to radiologic contrast dye | | Embarrassment | | |
| | None | Х | Possible anxiety or claustrophobia during MRI exam | | |
| | | | None | | |

c) Describe the procedures or safeguards in place to protect against or minimize potential risks (e.g., referral to psychological counseling resources).

-Standard assessment of allergy or MRI-associated risk prior to MRI study



| | A Data Safaty Manitoring Board (DSMR) State name of DSMR and describe procedures for | |
|---|---|---|
| | A Data Safety Monitoring Board (DSMB) State name of DSMB and describe procedures for submitting summary reports from the DSMB to the IRB: | |
| | Other: | |
| Are ther below as | attach DSMB reports. (see clinical research glossary for "DSMB" clarification. If you think your study warrants DSMB oversight and you do not know of one to utilize, please contact the IRB office.) e any stopping rules based on the risks noted above, or other study criteria? If yes, describe nd include study endpoints. (Click "Help" above for more information.)/ | N |
| | * * * Benefits * * * | |
| Benefits | (This section is not enabled for exempt or cooperative studies)/ | |
| Are ther outcome describe | e any direct benefits to the research participants? Note: Direct benefit is a valued or desired e; an advantage (please do not include monetary inducement or compensation). If yes, please e. | N |
| Are ther | e any anticipated benefits of this study to society, academic knowledge or both? If yes, please | Y |
| describe. The results of this study should define the effectiveness of MRI and/or CPK / aldolase as diagnostic tools in future patients with | | |
| | cted local anesthetic-induced myotoxicity | |
| Evolain | how the potential benefits justify the potential risks involved in participation in this research. | |
| LAPIGIII | | |



| | /MMC/BRI se<br>.ocked office | | X Investigator's com<br>N/A | ıputer | Locked file cabinet Other: (explain below) |
|---|---|---|---|---|---|
| e) | How will re | search records | be stored locally? | | |
| F | REDCap data<br>Other: ( | abase<br>explain below) | Patient medical re | ecords | N/A |
| d) | Case report f | search data be | Remote data entr | y (e.g. X<br>off site) | Local database (e.g. Excel spreadshee |
| -1\ | | | | | |
| | | (explain below) | Personal physicia | .11 ^ | None |
| | NIH<br>FDA | | Study Sponsor Personal physicia | ın V | Contracted monitor None |
| c) | Other than and/or data | study staff and<br>that identify su | BRI Regulatory & Com<br>bjects (including coded | pliance, what e<br>data)? | ntities will have access to research recor |
| | -CPK reports -A password- generated MI -MRNs will be | contain patient nan<br>protected spreadsh<br>RI standard reading<br>e removed from the | nes and medical record number<br>eet housed on a VMMC pass | bers, but will be see<br>sword-protected cor<br>with Dr. Steffel (at | en only by Dr. Neal and the patient's orthopedic tea<br>mputer will be used to link MRN to radiologist-<br>VA Puget Sound). |
| b) | Describe your protection method(s) in two or three sentences (e.g. coding system, limited access, password protected, certificate of confidentiality, etc.). Include safeguards to protect against direct or indirect identification of subjects in any reporting of research results (e.g. publications): -MRIs contain patient names and medical record numbers will be seen by the blinded radiologist | | | | |
| | Cod | ed | | | |
| | | nymous<br>dentified | | | |
| | | tifiable | | | |
| | • • | • | or more information)/ | | |

Describe in two or three sentences how the confidentiality of the retained information and/or specimens (whether directly identifiable or coded) will be maintained:



h) Indicate the length of time research records and/or specimens will be kept before EITHER all identifiers/codes are removed OR the records and/or specimens are destroyed. Describe the procedures you will use.

Research records will be kept 1 year after publication of our results. After that, the spreadsheet will be turned over to BRI for archiving.

\_\_\_\_\_

\* \* \* Consent Information \* \* \*

#### 12. Consent Information

Consent Instructions and Checklist
Template Consent Forms and Guidance

a) Click "Add" to enter information in the "Informed Consent" table below. This includes translated consents and waivers of consent. Exempt Studies: This table is disabled. If a consent is used then attach in the attachment section. Chart review: If accessing medical charts without consent, a waiver of consent is required. Oral Consent: A waiver of signed consent is required. Subjects under 18 yrs old: Go to the next section. complete and attach assent information. Enter information in the Informed Consent table separately for each consent and/or waiver of consent.

#### Informed Consent Table

| Title | Consent Type |
|-----------------------------------------------------------|--------------|
| Clean Consent - Vers. 04.09.18 - IRB18-008 | Consent |
| IRB Stamped Approved Consent - Vers. 04.09.18 - IRB18-008 | Consent |
| Revised Consent 5.17.18 | Consent |
| Consent 5.29.18 revision | Consent |

#### Informed Consent Table

Title (e.g. main, screening, translated, oral, information sheet, waiver request) \*

Clean Consent - Vers. 04.09.18 - IRB18-008

Consent Information Type\*

Consent

**Consent Document\*** 

X Attachment

Clean Consent - Vers. 04.09.18 -

IRB18-008

Who will obtain subjects consent? (Check all that apply)

**Principal Investigator** 

Co-Investigator

**Study Coordinator** 

Research assistant(s)

Other research staff

**Contracted Data Collection Firm** 

Other (please specify)

Informed Consent Table





Protocol: IRB18-008 PI Name: Neal, Joseph Date Printed: May 29, 2018

Title (e.g. main, screening, translated, oral,

information sheet, waiver request) \*

IRB Stamped Approved Consent - Vers. 04.09.18 - IRB18-008

**Consent Information Type\*** 

Consent

Χ

Consent Document\*

Attachment

IRB Stamped Approved Consent -Vers. 04.09.18 - IRB18-008

Who will obtain subjects consent? (Check all that apply)

**Principal Investigator** Х Co-Investigator

> **Study Coordinator** Research assistant(s) Other research staff

**Contracted Data Collection Firm** 

Other (please specify)

Informed Consent Table

Title (e.g. main, screening, translated, oral,

information sheet, waiver request) \*

Revised Consent 5.17.18

Attachment

Consent Information Type\*

**Consent Document\*** 

Consent Χ

Revised5.17.18.Consent Document -

Who will obtain subjects consent? (Check all that apply)

Х Principal Investigator

Χ Co-Investigator

> Study Coordinator Research assistant(s) Other research staff

**Contracted Data Collection Firm** 

Other (please specify)

Informed Consent Table

Title (e.g. main, screening, translated, oral,

information sheet, waiver request) \*

Consent 5.29.18 revision

Consent Information Type\*

Consent

**Consent Document\*** 

Х Attachment

IRB18-008 Consent Document.Rev

5.29.18

Who will obtain subjects consent? (Check all that apply)

Χ **Principal Investigator** Х

Co-Investigator

**Study Coordinator** Research assistant(s) Other research staff

**Contracted Data Collection Firm** 

Other (please specify)



If consenting human subjects answer the questions below. If NOT consenting human subjects, leave blank and skip to the next section. b) Describe the process used to consent all subjects on the study. -Volunteer subjects will be identified in orthopedic office by Dr. Verdin or his staff -Those interested in participating will be consented by Joseph M. Neal, MD at least 24 hours prior to their surgery. If possible, consent will be obtained in person. If not possible, consent will be obtained via phone. Will subjects have as much time as they want between the explanation of the study and signing the C) consent form? If no, or N/A explain below. d) If consent is being obtained from non-English speaking subjects, explain the translation process for all documents seen by subjects, including consent documents. Describe the consent process in these circumstances. N/A Do you plan on having a Legally Authorized Representative (LAR) involved in the consent process? If e) ves, explain below and ensure the appropriate section is included in the consent form. f) Will you require an impartial third party witness be included in the consenting process? If yes, explain below and ensure the appropriate section is included in the consent form. \* \* \* Assent Background \* \* \* Assent Background (Continue to the next section if no subjects under the age of 18 will be enrolled in this study) Complete the "Assent" table below. Attach assent documents and/or request assent waivers. Click "Help" above for more information regarding assent and assent waiver. You must check children (under 18) on the Subject Checklist section to activate this table. Complete the Regulatory Compliance worksheet below: Regulatory Compliance - Subpart D - Children Provide the specific age range for children (less than 18 years old) you wish to enroll in the study and what is your accrual goal: Age Range: Total Accrual Goal: Check the appropriate box below (only one) to indicate which category your study may be approved in light of 45 CFR 46 subpart D for research involving children. Chlick on the links below for guidance. Research not involving greater than minimal risk. 45 CFR 46.404 Research involving greater than minimal risk, but presenting the prospect of direct benefit to

the individual subjects. CFR 46.405



| | Research involving greater than minimal risk and no prospect of direct benefit to the individual child subjects involved in the research, but likely to yield generalizable knowledge about the subject's disorder or condition. 45 CFR 46.406 |
|---|---|
| | Research not otherwise approvable which presents an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of children. 45 CFR 46.407 |
| | Will you be using an Assent Form? (Required for subjects 7-11 years old per BRI IRB policies - see 45 CFR 46.408 for reference) |
| approach(es) to | space below the details of your assent process for children in your study. (Include specific subjects in various age ranges, how assent will be documented, who will be able to give each child (e.g. child's parent(s) or guardian), and how this permission will be recorded in the |
| | Does your study involve an FDA regulated drug, device, or biologic? If yes, check the appropriate box below (only one) to indicate which category your study may be approved in light of 21 CFR 50 Subpart D for research involving children. Click on the links below for guidance. |
| | Clinical investigations not involving greater than minimal risk 21 CFR 50.51 |
| | Clinical investigations involving greater than minimal risk, but presenting the prospect of direct benefit to the individual subjects. 21 CFR 50.52 |
| | Clinical investigations involving greater than minimal risk and no prospect of direct benefit to individual subjects. |
| | Clinical investigations not otherwise approvable that present an opportunity to understand, prevent, or alleviate a serious problem affecting the health or welfare of children. 21 CFR 50.53 |
| | Will you be using an Assent Form? (Required for subjects 7-11 years old per BRI IRB policies |

------

### \* \* \* HIPAA \* \* \*

14. Health Insurance Portability and Accountability Act (HIPAA)

- see 45 CFR 46.408 for reference)

If you are using PHI and this page is not active you must return to the General Checklist and check the box regarding the use of PHI in this research.

HIPAA Privacy Rule: Establishes the right of an individual to authorize a covered entity, such as health plan, health care clearinghouse or health care provider, to use and disclose his/her Protected Health Information (PHI) for research purposes. The Privacy Rule defines the elements of individual information that comprise PHI and establishes the conditions under which PHI may be used or disclosed by covered entities for research purposes. It also includes provisions to allow an individual's PHI to be disclosed or used in research without the person's authorization (i.e., IRB Waiver of HIPAA Requirement Authorization). For more information refer to the HIPAA Privacy Rule.

Protected Health Information (PHI):Health information with one or more of the identifiers listed below. For more information see the NIH website. Research which involves the use of de-identified data is exempt from HIPAA requirements. In order to be de-identified data NONE of the subject identifiers listed below can be collected, used, reviewed, recoded, accessed or disclosed.

For more information see the following:VM/BRI Protected Health Information Guidance Document

- a) How will you obtain approval to access PHI for this research?
  - X HIPAA Authorization request from subject
    - X Incorporated into consent form

Stand alone document



Waiver of Subject HIPAA Authorization (partial or complete)(complete question e. below) Limited Data Set and Data Use Agreement

Other: (explain below)

c) Will any non-VM/BRI personnel need access to PHI? If yes, how and where will they access subject PHI (e.g. on-site, remote via Cerner, etc.)?

Ν

d) Review the following list and indicate if any of the information will be collected from any medical records for the purpose of this research project.

**Names** 

**Social Security Numbers** 

**Telephone Numbers** 

All geographic subdivisions smaller than a state, including street address, city, county, precinct, zip code, and their equivalent geocodes, except for the initial three digits of a zip code, if according to the current publicly available data from the Bureau of the Census;

- i. The geographic unit formed by combining all zip codes with the same three initial digits contains more than 20,000 people; and
- ii. The initial three digits of a zip code for all such geographic units containing 20,000 or fewer people is changed to 000.

All elements of dates (except year) for dates directly related to an individual, including birth date, admission date, discharge date, date of death; and all ages over 89 and all elements of dates (including year) indicative of such age, except that such ages and elements may be aggregated into a single category of age 90 or older.

**Fax Numbers** 

Electronic Mail Addresses (email)

- X Medical Record Numbers
  - i. You must identify the data points being collected from MRN by attaching a separate data collection sheet or listing them in the procedures section.

**Health Plan Beneficiary Numbers** 

**Account Numbers** 

Certificate/License Numbers

Vehicle Identifiers and Serial Numbers, including License Plate Numbers

**Device Identifiers and Serial Numbers** 

Web Universal Resource Locations (URLs)

Internet Protocol (IP) Address Numbers

Biometric Identifiers, including Finger and Voice Prints

Full Face Photographic Images and any Comparable Images

Any other unique identifying number, character, or code (note this does not mean the unique code assigned by the Investigator(s) to code the research data)

| e) | Are you requesting a HIPAA waiver? | (Required for any type of waiver of consent)If yes, answer the |
|---|---|---|
| | following questions. If no, proceed to t | |

| Explain why the research cannot reasonably be conducted without the waiver of |
|---|
| authorization: |

Ν



| <br> | * * * Drugs and Devices * * * |
|---|---|
| | the research disclosures (e.g. PI, sub-investigator, coordinator): |
| viii. | Explain who the subject should contact to enforce patient rights, or to obtain an accounting of |
| vii. | Explain why the research is of sufficient importance to outweigh the privacy intrusion: |
| vi. | Provide written assurance that identifiable information will not be reused/disclosed to any other person or entity, unless such use is required by law, for oversight of the research study, or for other research permitted by law: |
| ٧. | research. If there is a health or research justification for retaining identifiers, or if law requires you to keep such identifying information, please provide this information as well: |
| v. | Describe the plan to destroy the identifiers at the earliest opportunity consistent with the |
| iv. | Describe the reasonable safeguards to protect against identification, directly or indirectly, any |
| iii. | Describe the reasonable safeguards to protect identifiable information from unauthorized use or re-disclosure: |
| | identifiable health information: |



- b) N If yes, are there any positive financial disclosures related to this study for any key personnel?
- c) N Regardless of funding, are there any positive positional disclosures related to this study for any key personnel?
- d) Y I attest that I have read the 
  'https://brinet.benaroyaresearch.org/center/Documents/VM%20Research%20Conflicts%20of%20Interes 
  t.pdf#search=research%20conflict'target='blank'VM Conflict of Interest Policy and agree to abide by its 
  terms. I will update this protocol when new or changes in conflict of interest arise, and I will comply with 
  any conflict management plan required by the Institutional Review Board (IRB) to manage, reduce, or 
  eliminate any actual or potential conflict of interest for the duration of the research.

If Yes to b) or c) above, complete the table and answer the questions below concerning the potential conflict of interest. If No, then proceed to the next section.

Minimizing Risks and Disclosure to Subjects

- N Have you disclosed any actual, potential or perceived conflicts of interest in the consent form? Research
  Personnel are required to disclose all such conflicts to all research participants in the research consent
  form.
- f) What steps, if any, have you taken or will you take to manage the conflict of interest and minimize the risks associated with any actual, potential or perceived conflicts of interest arising out of this research?

\_\_\_\_\_

\* \* \* Attachments \* \* \*

### 17. Attachments

Attach relevant documents here. These could include:

- Collaborating Investigator's IRB approval and approved documents
- Conflict of Interest information
- Debriefing Script; Grant/Sub-contract
- HIPAA Authorization Form from HIPAA-covered entity
- Interview/Focus Group Questions
- Investigator's Brochure
- Letters of Agreement/Cooperation from organizations who will help with recruitment
- Questionnaires/Surveys
- Radiation Control Office approval material
- Recruitment Material (e.g., flyers, email text, verbal scripts)
- Protocol
- Patient Card
- Other files associated with the protocol (you can upload most standard file formats: xls, pdf, jpg, tif, etc.)

Please be sure to attach all documents associated with your protocol. Failure to attach the necessary files may result in this protocol being returned prior to review.

To update or revise any attachments, please delete the existing attachment and upload the revised document to replace it.

| Select from list | Attachment Name | Attached Date | Submitted Date |
|------------------|-----------------|---------------|----------------|



| Data Collection Sheet | IRB18-008 Copy of Study<br>Data Sheet | 03/08/2018 | 05/22/2018 |
|---|---|---|---|
| Other | IRB18-008 Neal Financial Disclosure | 03/08/2018 | 05/22/2018 |
| Data Collection Sheet | IRB18-008 Copy of MRI<br>Data Sheet | 03/08/2018 | 05/22/2018 |
| Protocol | Clean Protocol - Vers.<br>04.09.18 - IRB18-008 | 04/13/2018 | 04/13/2018 |
| Protocol | IRB18-008 Protocol.Rev | 05/29/2018 | 05/29/2018 |

## \* \* \* Obligations \* \* \*

Note: The use of "I" below refers to the Principal Investigator (PI). If someone other than the PI is completing and submitting this application, that person is responsible to make sure the PI is aware of their obligation and assurances cited below. The PI is ultimately responsible for all conduct under this study and answers provided in this IRB submission.

#### Research Obligations of the Principal Investigator Include the Following:

5.29.18

Training - ALL key personnel, including any newly added personnel, must meet all IRB required training requirements (e.g. CITI Ethics, GCP, Conflict of Interest). Training refreshers must be completed at the appropriate intervals (i.e. every three (3) or four (4) years).

Study Modifications - Changes to any aspect of the study (e.g. protocol, consent/assent forms, advertising materials, additional key personnel, subject population, etc.) will be submitted to the IRB for approval before instituting the changes.

Final Report - The IRB will be notified when the study is complete, and must be closed out in eProtocol prior to expiration of the approval.

#### Investigator's Statement and Assurance of Confidentiality:

I certify that I have reviewed this application, including attachments, and all information contained herein is accurate to the best of my knowledge.

I agree to not enroll any subject(s) or collect any data intended only for research use prior to issuance of an IRB approval.

I understand that I am fully responsible for the execution and management of this study, and I am responsible for the performance of any sub-investigators or key personnel, including their adherence to all of the applicable policies and regulations.

I agree to report any substantive changes to the information contained in this application, unanticipated problems, or adverse events encountered during the project immediately to the IRB.

I will ensure the names of any human subjects or any identifiable data from human subjects shall be treated as confidential information. This information will not be disclosed to anyone other than those directly connected with the research project unless the patient has given prior approval in writing.

If this is a funded project, I certify that the funding source document is entirely consistent with the corresponding study protocol.

I certify I have not been barred from doing research by any regulatory agency or entity. If I am a physician (or other licensed health care professional), I certify that my medical (or other) license is current.

I further agree any failure to perform the undertaking specified above shall be good cause for termination of the research project.

### When Closing Your Protocol:

I understand when I close this protocol with the IRB NO further data collection, follow-up with subjects, coding of data, data analysis, and manuscript preparation that requires personal identifiable information (e.g. PHI) may be conducted.

I agree to retain all research materials for at least 10 years after closure of the research project and acknowledge these documents may be subject to review by the Clinical Research Program and IRB, if deemed necessary.

I further certify I will not take any PHI and/or specimens generated from this research with me if I leave BRI/VM, unless having first established an agreement with VM legal in advance of my departure.

### I confirm this study will not begin until the investigator receives written final approval or determination of exemption.

X The Principal Investigator has read and agrees to abide by the above obligations.





Continuing Review - You are responsible to complete and submit a Continuing Review form at least 30 days prior to the date of expiration. You will be asked to note accomplishments of your project at that time.

Protocol Deviations/Violations, Adverse Events (AEs) that occur in the course of the protocol will need to be submitted in a prompt manner from when they occurred.

X The Principal Investigator has read and agrees to abide by the above obligations.

Please click "next" to continue to protocol Check for Completeness. If the protocol is complete and ready for submission, please click "Submit Form" to your left to submit your protocol for IRB Review.

\_\_\_\_\_

## \* \* \* Event History \* \* \*

## **Event History**

| Date | Status | View Attachments | Letters |
|---|---|---|---|
| 05/29/2018 | AMENDMENT 2 FORM<br>SUBMITTED | Υ | |
| 05/29/2018 | AMENDMENT 2 FORM CREATED | | |
| 05/24/2018 | AMENDMENT 1 FORM<br>APPROVED | Υ | Y |
| 05/23/2018 | AMENDMENT 1 FORM REVIEWER(S) ASSIGNED | | |
| 05/22/2018 | AMENDMENT 1 FORM SUBMITTED | Υ | |
| 05/17/2018 | AMENDMENT 1 FORM CREATED | | |
| 04/30/2018 | NEW FORM APPROVED | Υ | Υ |
| 04/30/2018 | NEW FORM UNDO<br>APPROVED | | |
| 04/30/2018 | NEW FORM APPROVED | Υ | Υ |
| 04/17/2018 | NEW FORM REVIEWER(S) ASSIGNED | | |
| 04/13/2018 | NEW FORM REVIEWER(S) ASSIGNED | | |
| 04/12/2018 | NEW FORM PANEL<br>MANAGER REVIEW | | |
| 03/08/2018 | NEW FORM PANEL<br>ASSIGNED | | |
| 03/08/2018 | NEW FORM SUBMITTED | Υ | |
| 01/26/2018 | NEW FORM CREATED | | |